CLINICAL TRIAL: NCT02886728
Title: A Randomized, Double-blind, Placebo- and Active-controlled, Multicenter, Phase 3 Study to Assess the Efficacy and Safety of Filgotinib Administered for 52 Weeks Alone and in Combination With Methotrexate (MTX) to Subjects With Moderately to Severely Active Rheumatoid Arthritis Who Are Naïve to MTX Therapy
Brief Title: Filgotinib Alone and in Combination With Methotrexate (MTX) in Adults With Moderately to Severely Active Rheumatoid Arthritis Who Are Naive to MTX Therapy
Acronym: FINCH 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-417-0303; 2016-000570-37 (EudraCT Number)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Filgotinib 200 mg + MTX (Experimental): Filgotinib 200 mg + placebo to match filgotinib 100 mg + MTX up to 20 mg
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: MTX
- Filgotinib 100 mg + MTX (Experimental): Filgotinib 100 mg + placebo to match filgotinib 200 mg + MTX up to 20 mg
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: MTX
- Filgotinib 200 mg Monotherapy (Experimental): Filgotinib 200 mg + placebo to match filgotinib 100 mg + placebo to match MTX
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: Placebo to match MTX
- MTX Monotherapy (Active Comparator): Placebo to match filgotinib 200 mg + placebo to match filgotinib 100 mg + MTX up to 20 mg
  Interventions: Drug: Placebo to match filgotinib; Drug: MTX

INTERVENTIONS:
Drug: Filgotinib — Tablet(s) administered orally once daily
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib 100 mg + MTX; Filgotinib 200 mg + MTX; Filgotinib 200 mg Monotherapy
Drug: Placebo to match filgotinib — Tablet(s) administered orally once daily
Drug: MTX — Capsule(s) administered orally once weekly
  Arms: Filgotinib 100 mg + MTX; Filgotinib 200 mg + MTX; MTX Monotherapy
Drug: Placebo to match MTX — Capsule(s) administered orally once weekly
  Arms: Filgotinib 200 mg Monotherapy

SUMMARY:
The primary objective of this study is to evaluate the effects of filgotinib in combination with methotrexate (MTX) versus MTX alone in adults with active rheumatoid arthritis (RA).

ELIGIBILITY:
Key Inclusion Criteria:

* Have a diagnosis of RA (2010 American College of Rheumatology [ACR]/European League Against Rheumatism [EULAR] criteria) and are ACR functional class I-III.
* Have ≥ 6 swollen joints (from a swollen joint count based on 66 joints (SJC66)) and ≥ 6 tender joints (from a tender joint count based on 68 joints (TJC68)) at both screening and Day 1.
* Limited or no prior treatment with MTX

Key Exclusion Criteria:

* Previous treatment with any janus kinase (JAK) inhibitor
* Previous therapy for longer than 3 months with conventional synthetic disease modifying antirheumatic drugs (csDMARDs) other than MTX or hydroxychloroquine
* Use of any licensed or investigational biologic disease-modifying antirheumatic drugs (DMARDs)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1252 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (186):
- United States (45):
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Covina, California
  - Los Angeles, California
  - Palm Desert, California
  - Victorville, California
  - Whittier, California
  - DeBary, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Springfield, Illinois
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Cumberland, Maryland
  - Wheaton, Maryland
  - Worcester, Massachusetts
  - Saint Clair Shores, Michigan
  - Eagan, Minnesota
  - Hattiesburg, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Lebanon, New Hampshire
  - Freehold, New Jersey
  - Toms River, New Jersey
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bethlehem, Pennsylvania
  - Duncansville, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Orangeburg, South Carolina
  - Memphis, Tennessee
  - Beaumont, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Mesquite, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Webster, Texas
- Argentina (7):
  - Buenos Aires
  - Caba
  - Mendoza
  - Quilmes
  - San Fernando
  - San Juan
  - San Miguel de Tucumán
- Australia (3):
  - Maroochydore, Queensland
  - Hobart, Tasmania
  - Victoria Park, Western Australia
- Belgium (4):
  - Leuven, Flemish Brabant
  - Genk
  - Hasselt
  - Merksem
- Bulgaria (6):
  - Dobrich
  - Haskovo
  - Plovdiv
  - Sofia
  - Varna
  - Vidin
- Canada (2):
  - Barrie, Ontario
  - Trois-Rivières, Quebec
- Chile (2):
  - Santiago
  - Temuco
- Czechia (3):
  - Ostrava
  - Prague
  - Uherské Hradiště
- Germany (3):
  - Aachen
  - Hamburg
  - Ratingen
- Hong Kong (2):
  - Hong Kong
  - Tuenmen
- Hungary (4):
  - Kalocsa, Bács-Kiskun county
  - Székesfehérvár, Fejér
  - Budapest
  - Kistarcsa
- India (16):
  - Ahmedabad
  - Bangalore
  - Delhi
  - Jaipur
  - Kolkata
  - Lucknow
  - Mangalore
  - Mysuru
  - Nagpur
  - New Delhi
  - Pune
  - Secunderabad
  - Srikakulam
  - Surat
  - Vadodara
  - Visakhapatnam
- Dublin, Ireland
- Petah Tikva, Israel
- Italy (2):
  - Bologna
  - Reggio Emilia
- Japan (16):
  - Fukuoka
  - Hamamatsu
  - Hiroshima
  - Kagoshima
  - Katō
  - Kawagoe
  - Miyagi
  - Nagaoka
  - Nagasaki
  - Okayama
  - Ōme
  - Sanuki
  - Sapporo
  - Sasebo
  - Sayama
  - Tokyo
- Malaysia (2):
  - Batu Caves
  - Kuala Lumpur
- Mexico (6):
  - Mérida, Yucatán
  - Chihuahua City
  - Distrito Federal
  - Mérida
  - Monterrey
  - Morelia
- New Zealand (4):
  - Timaru, Canterbury
  - Hamilton
  - Newtown
  - Papatoetoe
- Poland (12):
  - Bialystok
  - Bydgoszcz
  - Bytom
  - Dąbrówka
  - Elblag
  - Gdynia
  - Katowice
  - Krakow
  - Nowa Sól
  - Poznan
  - Torun
  - Warsaw
- Romania (3):
  - Târgu Mureş, Mureș County
  - Bucharest
  - Oradea
- Russia (6):
  - Barnaul
  - Kemerovo
  - Moscow
  - Nizhny Novgorod
  - Saratov
  - Yaroslavl
- Belgrade, Serbia
- Slovakia (3):
  - Bratislava
  - Prievidza
  - Topoľčany
- South Africa (2):
  - Cape Town
  - Durban
- South Korea (5):
  - Anyang-si
  - Daegu
  - Daejeon
  - Incheon
  - Seoul
- Spain (7):
  - Sabadell, Barcelona
  - A Coruña
  - Barakaldo
  - Málaga
  - Sabadell
  - Santiago de Compostela
  - Valencia
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Songkhla
- Ukraine (8):
  - Dnipro
  - Kharkiv
  - Kherson
  - Kyiv
  - Lviv
  - Vinnitsa
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (2):
  - Edinburgh
  - Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Westhovens R, Rigby W, van der Heijde D, Ching D, Bartok B, Matzkies F, et al. Efficacy and safety of filgotinib for patients with rheumatoid arthritis naive to methotrexate therapy: FINCH 3 primary outcome results. Ann Rheum Dis 2019; 78 (supplement 2): A259.
- [Derived] Taylor PC, Downie B, Han L, Hawtin R, Hertz A, Moots RJ, Takeuchi T. Patients with High Baseline Neutrophil-to-Lymphocyte Ratio Exhibit Better Response to Filgotinib as Treatment for Rheumatoid Arthritis. Rheumatol Ther. 2024 Oct;11(5):1383-1392. doi: 10.1007/s40744-024-00695-w. Epub 2024 Jul 10. PMID 38985247
- [Derived] Curtis JR, Emery P, Downie B, Zhong Y, Liu J, Han L, Hawtin RE, Burmester GR. Filgotinib Demonstrates Efficacy in Rheumatoid Arthritis Independent of Smoking Status: Post Hoc Analysis of Phase 3 Trials and Claims-Based Analysis. Rheumatol Ther. 2024 Feb;11(1):177-189. doi: 10.1007/s40744-023-00619-0. Epub 2023 Dec 6. PMID 38057656
- [Derived] Balsa A, Wassenberg S, Tanaka Y, Tournadre A, Orzechowski HD, Rajendran V, Lendl U, Stiers PJ, Watson C, Caporali R, Galloway J, Verschueren P. Effect of Filgotinib on Body Mass Index (BMI) and Effect of Baseline BMI on the Efficacy and Safety of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Dec;10(6):1555-1574. doi: 10.1007/s40744-023-00599-1. Epub 2023 Sep 25. PMID 37747626
- [Derived] Tanaka Y, Atsumi T, Aletaha D, Bartok B, Pechonkina A, Han L, Emoto K, Kano S, Rajendran V, Takeuchi T. Benefit of Filgotinib, a JAK1 Preferential Inhibitor, in Rheumatoid Arthritis Patients with Previous Rapid Radiographic Progression: Post Hoc Analysis of Two Trials. Rheumatol Ther. 2023 Feb;10(1):161-185. doi: 10.1007/s40744-022-00503-3. Epub 2022 Nov 3. PMID 36327094
- [Derived] Combe B, Besuyen R, Gomez-Centeno A, Matsubara T, Sancho Jimenez JJ, Yin Z, Buch MH. Geographic Analysis of the Safety and Efficacy of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Feb;10(1):35-51. doi: 10.1007/s40744-022-00494-1. Epub 2022 Oct 7. PMID 36205910
- [Derived] Bingham CO 3rd, Walker D, Nash P, Lee SJ, Ye L, Hu H, Khalid JM, Combe B. The impact of filgotinib on patient-reported outcomes and health-related quality of life for patients with active rheumatoid arthritis: a post hoc analysis of Phase 3 studies. Arthritis Res Ther. 2022 Jan 3;24(1):11. doi: 10.1186/s13075-021-02677-7. PMID 34980223
- [Derived] Aletaha D, Westhovens R, Gaujoux-Viala C, Adami G, Matsumoto A, Bird P, Messina OD, Buch MH, Bartok B, Yin Z, Guo Y, Hendrikx T, Burmester GR. Efficacy and safety of filgotinib in methotrexate-naive patients with rheumatoid arthritis with poor prognostic factors: post hoc analysis of FINCH 3. RMD Open. 2021 Aug;7(2):e001621. doi: 10.1136/rmdopen-2021-001621. PMID 34385364
- [Derived] Westhovens R, Rigby WFC, van der Heijde D, Ching DWT, Stohl W, Kay J, Chopra A, Bartok B, Matzkies F, Yin Z, Guo Y, Tasset C, Sundy JS, Jahreis A, Mozaffarian N, Messina OD, Landewe RB, Atsumi T, Burmester GR. Filgotinib in combination with methotrexate or as monotherapy versus methotrexate monotherapy in patients with active rheumatoid arthritis and limited or no prior exposure to methotrexate: the phase 3, randomised controlled FINCH 3 trial. Ann Rheum Dis. 2021 Jun;80(6):727-738. doi: 10.1136/annrheumdis-2020-219213. Epub 2021 Jan 15. PMID 33452004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Asia, Africa, Australia, Europe, North America, and South America. The first participant was screened on 08 August 2016. The last study visit occurred on 08 May 2019.
Pre-assignment Details: 1855 participants were screened.
Groups:
- Filgotinib 200 mg + MTX: Participants were administered filgotinib 200 mg orally, once daily + placebo to match (PTM) filgotinib 100 mg orally, once daily + MTX up to 20 mg orally, once weekly for up to 54 weeks.
- Filgotinib 100 mg + MTX: Participants were administered filgotinib 100 mg orally, once daily + PTM filgotinib 200 mg orally, once daily + MTX up to 20 mg orally, once weekly for up to 54 weeks.
- Filgotinib 200 mg Monotherapy: Participants were administered filgotinib 200 mg orally, once daily + PTM filgotinib 100 mg orally, once daily + PTM MTX orally, once weekly for up to 54 weeks.
- MTX Monotherapy: Participants were administered PTM filgotinib 200 mg orally, once daily+ PTM filgotinib 100 mg orally, once daily + MTX up to 20 mg orally, once weekly for up to 56 weeks.
Period: Overall Study
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Started | 417 | 207 | 210 | 418
Completed | 345 | 175 | 174 | 331
Not Completed | 72 | 32 | 36 | 87
Not completed — Withdrew Consent | 31 | 13 | 11 | 47
Not completed — Lost to Follow-up | 12 | 6 | 13 | 12
Not completed — Adverse Event | 13 | 5 | 5 | 11
Not completed — Investigator's Discretion | 11 | 7 | 5 | 11
Not completed — Death | 3 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 4
Not completed — Non-Compliance with Study Drug | 1 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Randomized but Not Dosed | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy | Total
Number analyzed (Participants) | 416 | 207 | 210 | 416 | 1249
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13.8) | 54 (12.6) | 52 (13.9) | 53 (13.7) | 53 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 325 | 158 | 166 | 312 | 961
  Male | 91 | 49 | 44 | 104 | 288
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    Race: American Indian or Alaska Native | 26 | 12 | 18 | 33 | 89
    Race: Asian: Japanese | 23 | 11 | 12 | 25 | 71
    Race: Asian: Chinese/Taiwanese/Hong Kong Chinese | 7 | 4 | 6 | 10 | 27
    Race: Asian: Vietnamese | 1 | 0 | 0 | 0 | 1
    Race: Asian: Korean | 6 | 8 | 2 | 8 | 24
    Race: Asian: Other | 53 | 28 | 27 | 42 | 150
    Race: Black or African American | 15 | 8 | 8 | 14 | 45
    Race: Native Hawaiian or Pacific Islander | 1 | 0 | 1 | 3 | 5
    Race: White | 278 | 132 | 135 | 278 | 823
    Race: Other | 6 | 4 | 0 | 3 | 13
    Race: Not Permitted | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 93 | 40 | 45 | 84 | 262
    Ethnicity: Not Hispanic or Latino | 322 | 167 | 165 | 332 | 986
    Ethnicity: Not Permitted | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112 | 47 | 54 | 106 | 319
  Spain | 12 | 5 | 7 | 10 | 34
  Germany | 7 | 7 | 6 | 10 | 30
  South Korea | 6 | 8 | 2 | 8 | 24
  Canada | 5 | 5 | 4 | 6 | 20
  Belgium | 3 | 2 | 6 | 8 | 19
  South Africa | 8 | 5 | 1 | 5 | 19
  Australia | 7 | 2 | 2 | 7 | 18
  New Zealand | 9 | 3 | 0 | 4 | 16
  United Kingdom | 1 | 1 | 1 | 5 | 8
  Italy | 2 | 0 | 1 | 0 | 3
  Ireland | 1 | 0 | 0 | 1 | 2
  Israel | 0 | 0 | 2 | 0 | 2
  India | 41 | 21 | 22 | 31 | 115
  Poland | 35 | 21 | 15 | 37 | 108
  Ukraine | 21 | 10 | 13 | 25 | 69
  Bulgaria | 17 | 11 | 8 | 18 | 54
  Russia | 9 | 4 | 4 | 14 | 31
  Czechia | 5 | 3 | 3 | 9 | 20
  Hungary | 7 | 2 | 3 | 6 | 18
  Serbia | 6 | 2 | 4 | 4 | 16
  Romania | 4 | 1 | 2 | 3 | 10
  Slovakia | 4 | 0 | 2 | 2 | 8
  Mexico | 35 | 20 | 23 | 38 | 116
  Argentina | 16 | 5 | 4 | 15 | 40
  Chile | 7 | 3 | 1 | 3 | 14
  Taiwan | 7 | 2 | 5 | 9 | 23
  Thailand | 5 | 2 | 1 | 5 | 13
  Malaysia | 1 | 3 | 1 | 1 | 6
  Hong Kong | 0 | 1 | 1 | 1 | 3
  Japan | 23 | 11 | 12 | 25 | 71

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20% Improvement (ACR20) Response at Week 24
Description: ACR20 response is achieved when the participant has: ≥ 20% improvement (reduction) from baseline in tender joint count based on 68 joints (TJC68), swollen joint count based on 66 joints (SJC66) and in at least 3 of the following 5 items: physician's global assessment of disease activity (PGA) and subject's global assessment of disease activity (SGA) assessed using visual analog scale (VAS) on a scale of 0-100 (0 and 100 indicating no disease activity and maximum disease activity); subject's pain assessment using VAS on a scale of 0-100 (0 and 100 indicating no pain and unbearable pain); health assessment questionnaire-disability index (HAQ-DI) score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 (0 and 3 indicating without difficulty and unable to do); high-sensitivity C-reactive protein (hsCRP). Participants with missing outcomes were set as non-responders.
Time Frame: Week 24
Population: The Full Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of participants | 81.0 [77.1 to 84.9] | 80.2 [74.5 to 85.9] | 78.1 [72.3 to 83.9] | 71.4 [66.9 to 75.9]
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 9.6, 95% CI 2-sided [3.6 to 15.6]
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p = 0.017, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 8.8, 95% CI 2-sided [1.5 to 16.1]
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24; Test type: Superiority; p = 0.058, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 6.7, 95% CI 2-sided [-0.7 to 14.1]

2. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0-3 [0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices]. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0-3 [0 (no disability) to 3 (completely disabled)] when 6 or more categories are non-missing, total possible score is 3. If more than 2 categories are missing, the HAQ-DI score is set to missing. Negative change from baseline indicates improvement (less disability).
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 414 | 207 | 210 | 416
  Baseline | 1.52 (0.622) | 1.56 (0.654) | 1.56 (0.655) | 1.60 (0.625)
  Change at Week 24: number analyzed (Participants) | 372 | 190 | 185 | 370
  Change at Week 24 | -0.94 (0.722) | -0.90 (0.675) | -0.89 (0.631) | -0.79 (0.634)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24. LS-Mean, 95% CI, and P-value were provided from mixed effects model for repeated measures (MMRM). Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — MMRM model included treatment, visit, treatment by visit, stratification factors, and baseline value as fixed effects, and participants being the random effect; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-0.27 to -0.11], Standard Error of Mean 0.041
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.009, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.13, 95% CI 2-sided [-0.23 to -0.03], Standard Error of Mean 0.049
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.032, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.11, 95% CI 2-sided [-0.20 to -0.01], Standard Error of Mean 0.050

3. Secondary Outcome: Percentage of Participants Who Achieved Disease Activity Score for 28 Joint Count Using C-Reactive Protein [DAS28 (CRP)] < 2.6 at Week 24
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), Patient's Global Assessment of Disease Activity (visual analog scale: 0 = no disease activity to 100 = maximum disease activity), and CRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. Participants with missing outcomes were set as non-responders.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of participants | 54.1 [49.2 to 59.0] | 42.5 [35.5 to 49.5] | 42.4 [35.5 to 49.3] | 29.1 [24.6 to 33.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 25.0, 95% CI 2-sided [18.3 to 31.7]
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.4, 95% CI 2-sided [5.0 to 21.8]
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.3, 95% CI 2-sided [5.0 to 21.6]

4. Secondary Outcome: Change From Baseline in the Modified Total Sharp Score (mTSS) at Week 24
Description: Participant's radiographs of bilateral hands, wrists and feet are taken and evaluated through central review using the mTSS method. The mTSS (range [0-448]) is defined as the erosion score (range [0-280]) plus the joint space narrowing (JSN) score (range [0-168]). An erosion score of 0 to 5 is given to each joint in the hands and wrists, and a score of 0 to 10 is given to each joint in the feet [where 0 indicates no erosion while 5 or 10 indicates extensive loss of bone (maximum erosion]). JSN is scored from 0 to 4 [0 indicating no/normal JSN and 4 indicating complete loss of joint space]. The maximal TSS is 448. Positive change in value indicates progression of disease (more erosion of bone, less joint spaces).
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 410 | 204 | 204 | 408
  Baseline | 11.35 (19.922) | 13.31 (26.980) | 16.53 (32.372) | 13.72 (29.168)
  Change at Week 24: number analyzed (Participants) | 355 | 184 | 173 | 356
  Change at Week 24 | 0.21 (1.684) | 0.22 (1.526) | -0.04 (1.710) | 0.51 (2.887)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.068, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.29, 95% CI 2-sided [-0.61 to 0.02], Standard Error of Mean 0.161
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.14, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.29, 95% CI 2-sided [-0.67 to 0.10], Standard Error of Mean 0.195
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.55, 95% CI 2-sided [-0.94 to -0.16], Standard Error of Mean 0.199

5. Secondary Outcome: Change From Baseline in 36-Item Short Form Survey (SF-36) Physical Component Summary (PCS) Score at Week 24
Description: The SF-36 is a 36-item, self-reported, generic, comprehensive, and health-related quality of life questionnaire based on 8 health domains in 2 components: physical well-being (physical functioning, role-physical, bodily pain, general health perceptions), mental well-being (vitality, social functioning, role-emotional, and mental health). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with highest possible score of 100. Higher scores indicate better health status or functioning. Positive change in value indicates improvement and better quality of life.
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 414 | 207 | 208 | 416
  Baseline | 33.9 (7.48) | 33.7 (8.00) | 33.6 (7.70) | 33.3 (7.28)
  Change at Week 24: number analyzed (Participants) | 373 | 190 | 185 | 371
  Change at Week 24 | 12.3 (8.89) | 11.1 (9.00) | 10.4 (9.09) | 9.7 (8.62)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.9, 95% CI 2-sided [1.8 to 4.0], Standard Error of Mean 0.56
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.021, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.6, 95% CI 2-sided [0.2 to 2.9], Standard Error of Mean 0.69
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.24, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.8, 95% CI 2-sided [-0.5 to 2.2], Standard Error of Mean 0.69

6. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 24
Description: FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scales for a total possible score of 52. Positive change in value indicates improvement (no or less severity of fatigue).
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 411 | 207 | 206 | 415
  Baseline | 28.3 (10.93) | 27.3 (11.92) | 27.3 (10.90) | 27.1 (10.72)
  Change at Week 24: number analyzed (Participants) | 365 | 189 | 181 | 365
  Change at Week 24 | 10.6 (11.49) | 11.4 (11.26) | 10.2 (11.37) | 10.1 (11.19)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.056, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.3, 95% CI 2-sided [-0.0 to 2.6], Standard Error of Mean 0.68
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.10, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.3, 95% CI 2-sided [-0.3 to 3.0], Standard Error of Mean 0.82
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.67, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.4, 95% CI 2-sided [-1.3 to 2.0], Standard Error of Mean 0.83

7. Secondary Outcome: Change From Baseline in the mTSS at Week 52
Description: as for outcome 4
Time Frame: Baseline; Week 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 411 | 205 | 204 | 408
  Baseline | 11.31 (19.273) | 12.76 (24.363) | 15.89 (31.813) | 13.36 (27.736)
  Change at Week 52: number analyzed (Participants) | 345 | 176 | 166 | 330
  Change at Week 52 | 0.31 (1.808) | 0.23 (1.111) | 0.33 (1.902) | 0.81 (3.089)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — MMRM model included treatment, visit, treatment by visit, stratification factors, campaign groups, and baseline value as fixed effects, and participants being the random effect; Least Squares Mean Difference = -0.65, 95% CI 2-sided [-1.03 to -0.27], Standard Error of Mean 0.195
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.008, MMRM — [p-value comment as in outcome 7, analysis 1]; Least Squares Mean Difference = -0.63, 95% CI 2-sided [-1.09 to -0.16], Standard Error of Mean 0.236
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 7, analysis 1]; Least Squares Mean Difference = -0.66, 95% CI 2-sided [-1.14 to -0.19], Standard Error of Mean 0.242

8. Secondary Outcome: Percentage of Participants Who Achieved ACR20 Response at Weeks 2, 4, 12, 36, and 52
Description: ACR20 response is achieved when the participant has: ≥ 20% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions,8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 12, 36, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of participants
  Week 2 | 42.1 [37.2 to 46.9] | 37.2 [30.4 to 44.0] | 39.5 [32.7 to 46.4] | 16.6 [12.9 to 20.3]
  Week 4 | 62.3 [57.5 to 67.0] | 55.6 [48.5 to 62.6] | 52.4 [45.4 to 59.4] | 33.4 [28.8 to 38.1]
  Week 12 | 76.7 [72.5 to 80.9] | 72.0 [65.6 to 78.3] | 71.4 [65.1 to 77.8] | 59.4 [54.5 to 64.2]
  Week 36 | 75.5 [71.2 to 79.7] | 73.4 [67.2 to 79.7] | 76.2 [70.2 to 82.2] | 68.3 [63.7 to 72.9]
  Week 52 | 75.0 [70.7 to 79.3] | 73.4 [67.2 to 79.7] | 74.8 [68.6 to 80.9] | 61.8 [57.0 to 66.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 25.5, 95% CI 2-sided [19.3 to 31.7]
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 20.6, 95% CI 2-sided [12.8 to 28.5]
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 22.9, 95% CI 2-sided [15.1 to 30.8]
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 28.8, 95% CI 2-sided [22.1 to 35.6]
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 22.1, 95% CI 2-sided [13.6 to 30.7]
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.0, 95% CI 2-sided [10.5 to 27.5]
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 17.3, 95% CI 2-sided [10.8 to 23.8]
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p = 0.002, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.6, 95% CI 2-sided [4.5 to 20.7]
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 12; Test type: Superiority; p = 0.002, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.1, 95% CI 2-sided [4.0 to 20.1]
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.016, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.2, 95% CI 2-sided [0.9 to 13.5]
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.18, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 5.2, 95% CI 2-sided [-2.7 to 13.0]
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.030, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.9, 95% CI 2-sided [0.3 to 15.6]
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.2, 95% CI 2-sided [6.7 to 19.7]
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p = 0.003, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.7, 95% CI 2-sided [3.7 to 19.6]
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.0, 95% CI 2-sided [5.1 to 20.8]

9. Secondary Outcome: Percentage of Participants Who Achieved ACR 50% Improvement (ACR50) at Weeks 2, 4, 12, 24, 36, and 52
Description: ACR50 response is achieved when the participant has: ≥ 50% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions,8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of participants
  Week 2 | 13.0 [9.6 to 16.3] | 9.2 [5.0 to 13.4] | 16.2 [11.0 to 21.4] | 2.9 [1.2 to 4.6]
  Week 4 | 29.3 [24.8 to 33.8] | 20.8 [15.0 to 26.5] | 25.7 [19.6 to 31.9] | 9.4 [6.5 to 12.3]
  Week 12 | 53.1 [48.2 to 58.0] | 44.4 [37.4 to 51.5] | 45.7 [38.7 to 52.7] | 28.4 [23.9 to 32.8]
  Week 24 | 61.5 [56.7 to 66.3] | 57.0 [50.0 to 64.0] | 58.1 [51.2 to 65.0] | 45.7 [40.8 to 50.6]
  Week 36 | 60.6 [55.8 to 65.4] | 55.6 [48.5 to 62.6] | 58.6 [51.7 to 65.5] | 48.6 [43.6 to 53.5]
  Week 52 | 62.3 [57.5 to 67.0] | 59.4 [52.5 to 66.4] | 61.4 [54.6 to 68.3] | 48.3 [43.4 to 53.2]
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 10.1, 95% CI 2-sided [6.2 to 13.9]
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p = 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 6.3, 95% CI 2-sided [1.7 to 10.9]
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.3, 95% CI 2-sided [7.7 to 18.9]
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 20.0, 95% CI 2-sided [14.5 to 25.4]
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.4, 95% CI 2-sided [4.8 to 18.0]
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.3, 95% CI 2-sided [9.4 to 23.2]
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 24.8, 95% CI 2-sided [18.1 to 31.5]
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.1, 95% CI 2-sided [7.7 to 24.5]
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 17.3, 95% CI 2-sided [9.0 to 25.7]
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 15.9, 95% CI 2-sided [8.9 to 22.8]
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p = 0.006, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.3, 95% CI 2-sided [2.7 to 20.0]
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24; Test type: Superiority; p = 0.002, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.4, 95% CI 2-sided [3.9 to 21.0]
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.0, 95% CI 2-sided [5.1 to 19.0]
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.090, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.0, 95% CI 2-sided [-1.7 to 15.7]
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.014, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 10.0, 95% CI 2-sided [1.4 to 18.6]
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.9, 95% CI 2-sided [7.0 to 20.9]
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p = 0.008, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.1, 95% CI 2-sided [2.5 to 19.7]
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52; Test type: Superiority; p = 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.1, 95% CI 2-sided [4.6 to 21.6]

10. Secondary Outcome: Percentage of Participants Who Achieved ACR 70% Improvement (ACR70) at Weeks 2, 4, 12, 24, 36, and 52
Description: ACR70 response is achieved when the participant has: ≥ 70% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions,8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of participants
  Week 2 | 3.1 [1.3 to 4.9] | 1.9 [0.0 to 4.0] | 4.3 [1.3 to 7.3] | 0.7 [0.0 to 1.7]
  Week 4 | 13.0 [9.6 to 16.3] | 6.3 [2.7 to 9.8] | 11.4 [6.9 to 16.0] | 3.8 [1.9 to 5.8]
  Week 12 | 32.9 [28.3 to 37.6] | 27.1 [20.8 to 33.3] | 29.0 [22.7 to 35.4] | 13.2 [9.8 to 16.6]
  Week 24 | 43.8 [38.9 to 48.6] | 40.1 [33.2 to 47.0] | 40.0 [33.1 to 46.9] | 26.0 [21.6 to 30.3]
  Week 36 | 45.9 [41.0 to 50.8] | 37.2 [30.4 to 44.0] | 39.5 [32.7 to 46.4] | 32.2 [27.6 to 36.8]
  Week 52 | 47.8 [42.9 to 52.8] | 40.1 [33.2 to 47.0] | 45.2 [38.3 to 52.2] | 29.8 [25.3 to 34.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p = 0.018, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 2.4, 95% CI 2-sided [0.3 to 4.5]
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p = 0.17, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 1.2, 95% CI 2-sided [-1.2 to 3.6]
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 2; Test type: Superiority; p = 0.004, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 3.6, 95% CI 2-sided [0.3 to 6.8]
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 9.1, 95% CI 2-sided [5.2 to 13.1]
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p = 0.18, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 2.4, 95% CI 2-sided [-1.7 to 6.6]
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.6, 95% CI 2-sided [2.5 to 12.6]
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.7, 95% CI 2-sided [13.9 to 25.5]
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.8, 95% CI 2-sided [6.6 to 21.1]
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 15.8, 95% CI 2-sided [8.5 to 23.1]
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 17.8, 95% CI 2-sided [11.2 to 24.4]
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.1, 95% CI 2-sided [5.9 to 22.4]
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.0, 95% CI 2-sided [5.8 to 22.2]
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.7, 95% CI 2-sided [6.9 to 20.5]
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.20, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 5.0, 95% CI 2-sided [-3.3 to 13.3]
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.056, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.3, 95% CI 2-sided [-1.0 to 15.7]
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.0, 95% CI 2-sided [11.3 to 24.8]
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p = 0.010, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 10.3, 95% CI 2-sided [1.9 to 18.6]
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 15.4, 95% CI 2-sided [7.0 to 23.8]

11. Secondary Outcome: Change From Baseline in Individual ACR Component: HAQ-DI at Weeks 2, 4, 12, 36, and 52
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled). A negative change from baseline indicates improvement (less disability).
Time Frame: Baseline; Weeks 2, 4, 12, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 414 | 207 | 210 | 416
  Baseline | 1.52 (0.622) | 1.56 (0.654) | 1.56 (0.655) | 1.60 (0.625)
  Change at Week 2: number analyzed (Participants) | 400 | 202 | 202 | 405
  Change at Week 2 | -0.37 (0.495) | -0.36 (0.490) | -0.32 (0.442) | -0.18 (0.426)
  Change at Week 4: number analyzed (Participants) | 405 | 200 | 205 | 403
  Change at Week 4 | -0.57 (0.587) | -0.45 (0.547) | -0.51 (0.526) | -0.32 (0.511)
  Change at Week 12: number analyzed (Participants) | 389 | 197 | 193 | 389
  Change at Week 12 | -0.85 (0.698) | -0.77 (0.670) | -0.76 (0.625) | -0.61 (0.582)
  Change at Week 36: number analyzed (Participants) | 348 | 178 | 179 | 327
  Change at Week 36 | -0.96 (0.725) | -0.93 (0.700) | -0.91 (0.673) | -0.89 (0.675)
  Change at Week 52: number analyzed (Participants) | 332 | 169 | 171 | 307
  Change at Week 52 | -1.00 (0.728) | -0.97 (0.719) | -0.95 (0.688) | -0.88 (0.685)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 2. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — MMRM model included treatment, visit, treatment by visit, stratification factors, and baseline value as fixed effects, and subjects being the random effect; Least Squares Mean Difference = -0.23, 95% CI 2-sided [-0.29 to -0.17], Standard Error of Mean 0.031
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 2. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.20, 95% CI 2-sided [-0.28 to -0.13], Standard Error of Mean 0.038
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 2. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.17, 95% CI 2-sided [-0.24 to -0.09], Standard Error of Mean 0.038
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 4. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.29, 95% CI 2-sided [-0.35 to -0.22], Standard Error of Mean 0.035
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 4. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.15, 95% CI 2-sided [-0.23 to -0.06], Standard Error of Mean 0.043
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 4. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.21, 95% CI 2-sided [-0.29 to -0.12], Standard Error of Mean 0.042
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 12. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.28, 95% CI 2-sided [-0.35 to -0.20], Standard Error of Mean 0.039
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 12. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.18, 95% CI 2-sided [-0.28 to -0.09], Standard Error of Mean 0.048
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 12. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.17, 95% CI 2-sided [-0.26 to -0.07], Standard Error of Mean 0.048
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 36. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.13, 95% CI 2-sided [-0.22 to -0.05], Standard Error of Mean 0.043
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 36. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.23, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.06, 95% CI 2-sided [-0.17 to 0.04], Standard Error of Mean 0.052
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 36. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.24, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.06, 95% CI 2-sided [-0.16 to 0.04], Standard Error of Mean 0.052
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.17, 95% CI 2-sided [-0.25 to -0.08], Standard Error of Mean 0.045
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.077, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.10, 95% CI 2-sided [-0.20 to 0.01], Standard Error of Mean 0.054
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.039, MMRM — [p-value comment as in outcome 11, analysis 1]; Least Squares Mean Difference = -0.11, 95% CI 2-sided [-0.22 to -0.01], Standard Error of Mean 0.054

12. Secondary Outcome: Change From Baseline in Individual ACR Component: Tender Joint Count Based on 68 Joints (TJC68) at Weeks 2, 4, 12, 24, 36, and 52
Description: TJC was examined on 68 joints of the fingers, elbows, hips, knees, ankles, and toes distal for pain in response to pressure or passive motion at the study time points. Joint pain was scored as 0 = Absent; 1 = Present for each joint. The overall Tender Joint Count ranged from 0 to 68. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
tender joint count
  Baseline | 26 (14.5) | 25 (13.9) | 26 (13.7) | 26 (13.8)
  Change at Week 2: number analyzed (Participants) | 402 | 202 | 201 | 405
  Change at Week 2 | -9 (10.2) | -8 (9.8) | -9 (11.2) | -5 (9.8)
  Change at Week 4: number analyzed (Participants) | 408 | 201 | 205 | 404
  Change at Week 4 | -13 (12.1) | -12 (10.1) | -13 (11.8) | -8 (11.5)
  Change at Week 12: number analyzed (Participants) | 390 | 197 | 193 | 387
  Change at Week 12 | -18 (12.5) | -17 (12.4) | -18 (12.4) | -15 (12.2)
  Change at Week 24: number analyzed (Participants) | 374 | 190 | 186 | 370
  Change at Week 24 | -20 (12.5) | -20 (13.0) | -22 (12.4) | -19 (12.9)
  Change at Week 36: number analyzed (Participants) | 348 | 178 | 179 | 327
  Change at Week 36 | -21 (12.6) | -21 (12.8) | -23 (11.9) | -21 (12.7)
  Change at Week 52: number analyzed (Participants) | 332 | 170 | 171 | 307
  Change at Week 52 | -22 (12.4) | -21 (13.0) | -23 (12.3) | -21 (12.6)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-6.0 to -3.0], Standard Error of Mean 0.8
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-6.0 to -2.0], Standard Error of Mean 0.9
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-7.0 to -3.0], Standard Error of Mean 0.9
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-7.0 to -4.0], Standard Error of Mean 0.7
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-6.0 to -3.0], Standard Error of Mean 0.9
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-7.0 to -3.0], Standard Error of Mean 0.9
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-5.0 to -2.0], Standard Error of Mean 0.7
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-5.0 to -2.0], Standard Error of Mean 0.8
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-6.0 to -2.0], Standard Error of Mean 0.8
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.5
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.005, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.6
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -1.0], Standard Error of Mean 0.6
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p = 0.063, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.0 to 0.0], Standard Error of Mean 0.5
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.64, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.0, 95% CI 2-sided [-1.0 to 1.0], Standard Error of Mean 0.6
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.6
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.5
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.095, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.0 to 0.0], Standard Error of Mean 0.6
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.6

13. Secondary Outcome: Change From Baseline in Individual ACR Component: Swollen Joint Count Based on 66 Joints (SJC66) at Weeks 2, 4, 12, 24, 36, and 52
Description: The total SJC66 was based on 66 joints (same 68 joints counted in TJC68 minus hips). It was derived as the sum of all "1s" thus collected with no penalty considered for the joints not assessed or those which had been replaced. The range for SJC66 is 0 to 66. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
swollen joint count
  Baseline | 16.0 (9.8) | 16.0 (9.3) | 16.0 (9.7) | 16.0 (9.4)
  Change at Week 2: number analyzed (Participants) | 402 | 202 | 201 | 405
  Change at Week 2 | -7.0 (8.0) | -6.0 (6.9) | -7.0 (8.1) | -4.0 (7.5)
  Change at Week 4: number analyzed (Participants) | 408 | 201 | 205 | 404
  Change at Week 4 | -9.0 (8.7) | -9.0 (7.6) | -9.0 (8.3) | -6.0 (9.2)
  Change at Week 12: number analyzed (Participants) | 390 | 197 | 193 | 387
  Change at Week 12 | -13.0 (8.9) | -12.0 (8.1) | -13.0 (9.1) | -11.0 (8.9)
  Change at Week 24: number analyzed (Participants) | 374 | 190 | 186 | 370
  Change at Week 24 | -14.0 (8.9) | -14.0 (8.8) | -15.0 (9.5) | -13.0 (8.8)
  Change at Week 36: number analyzed (Participants) | 348 | 178 | 179 | 327
  Change at Week 36 | -14.0 (9.1) | -14.0 (9.4) | -15.0 (9.7) | -14.0 (8.7)
  Change at Week 52: number analyzed (Participants) | 332 | 170 | 171 | 307
  Change at Week 52 | -15.0 (9.2) | -14.0 (8.9) | -16.0 (9.8) | -14.0 (9.0)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.7
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -1.0], Standard Error of Mean 0.7
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, Mixed effects model for repeated measure — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -2.0], Standard Error of Mean 0.5
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -1.0], Standard Error of Mean 0.6
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -1.0], Standard Error of Mean 0.6
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -2.0], Standard Error of Mean 0.4
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.5
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-4.0 to -2.0], Standard Error of Mean 0.5
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-2.0 to -1.0], Standard Error of Mean 0.3
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-2.0 to -1.0], Standard Error of Mean 0.4
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-3.0 to -1.0], Standard Error of Mean 0.4
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-1.0 to -0.0], Standard Error of Mean 0.2
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.12, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.0, 95% CI 2-sided [-1.0 to 0.0], Standard Error of Mean 0.3
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.019, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-1.0 to -0.0], Standard Error of Mean 0.3
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.0 to -1.0], Standard Error of Mean 0.2
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.032, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-1.0 to -0.0], Standard Error of Mean 0.3
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.0 to -0.0], Standard Error of Mean 0.3

14. Secondary Outcome: Change From Baseline in Individual ACR Component: Subject's Global Assessment of Disease Activity (SGA) at Weeks 2, 4, 12, 24, 36, and 52
Description: SGA was assessed by the participant using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline | 65.0 (21.0) | 66.0 (21.6) | 68.0 (19.2) | 66.0 (21.0)
  Change at Week 2: number analyzed (Participants) | 401 | 201 | 202 | 407
  Change at Week 2 | -17.0 (20.8) | -13.0 (18.9) | -14.0 (20.7) | -7.0 (18.9)
  Change at Week 4: number analyzed (Participants) | 407 | 200 | 205 | 404
  Change at Week 4 | -26.0 (24.7) | -20.0 (22.5) | -22.0 (24.6) | -14.0 (22.2)
  Change at Week 12: number analyzed (Participants) | 391 | 196 | 192 | 389
  Change at Week 12 | -37.0 (26.7) | -30.0 (26.1) | -32.0 (27.7) | -25.0 (25.9)
  Change at Week 24: number analyzed (Participants) | 374 | 190 | 184 | 370
  Change at Week 24 | -42.0 (26.8) | -36.0 (27.4) | -38.0 (26.6) | -34.0 (27.4)
  Change at Week 36: number analyzed (Participants) | 348 | 178 | 179 | 327
  Change at Week 36 | -43.0 (27.2) | -39.0 (27.8) | -39.0 (24.3) | -38.0 (28.0)
  Change at Week 52: number analyzed (Participants) | 332 | 170 | 171 | 307
  Change at Week 52 | -45.0 (27.0) | -41.0 (28.1) | -43.0 (25.4) | -38.0 (28.3)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -11.0, 95% CI 2-sided [-13.0 to -8.0], Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-10.0 to -4.0], Standard Error of Mean 1.6
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-10.0 to -3.0], Standard Error of Mean 1.6
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -12.0, 95% CI 2-sided [-15.0 to -10.0], Standard Error of Mean 1.5
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-10.0 to -2.0], Standard Error of Mean 1.8
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-11.0 to -4.0], Standard Error of Mean 1.8
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -12.0, 95% CI 2-sided [-15.0 to -9.0], Standard Error of Mean 1.6
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p = 0.009, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-9.0 to -1.0], Standard Error of Mean 2.0
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-10.0 to -2.0], Standard Error of Mean 2.0
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-13.0 to -6.0], Standard Error of Mean 1.6
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.11, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-7.0 to 1.0], Standard Error of Mean 2.0
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.066, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-8.0 to 0.0], Standard Error of Mean 2.0
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-11.0 to -4.0], Standard Error of Mean 1.7
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.40, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-6.0 to 2.0], Standard Error of Mean 2.1
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.24, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-6.0 to 2.0], Standard Error of Mean 2.1
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-12.0 to -5.0], Standard Error of Mean 1.7
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.17, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-7.0 to 1.0], Standard Error of Mean 2.1
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.008, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-10.0 to -1.0], Standard Error of Mean 2.1

15. Secondary Outcome: Change From Baseline in Individual ACR Component: Physician's Global Assessment of Disease Activity (PGA) at Weeks 2, 4, 12, 24, 36, and 52
Description: PGA was assessed by the physician using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline | 66.0 (17.0) | 68.0 (16.3) | 66.0 (14.4) | 67.0 (16.8)
  Change at Week 2: number analyzed (Participants) | 397 | 200 | 201 | 401
  Change at Week 2 | -24.0 (20.3) | -21.0 (19.4) | -23.0 (19.9) | -15.0 (18.9)
  Change at Week 4: number analyzed (Participants) | 402 | 201 | 198 | 402
  Change at Week 4 | -34.0 (22.3) | -32.0 (22.5) | -30.0 (21.9) | -23.0 (20.7)
  Change at Week 12: number analyzed (Participants) | 388 | 196 | 192 | 385
  Change at Week 12 | -47.0 (21.4) | -43.0 (22.5) | -42.0 (20.8) | -38.0 (21.9)
  Change at Week 24: number analyzed (Participants) | 372 | 187 | 185 | 364
  Change at Week 24 | -51.0 (21.1) | -51.0 (22.2) | -49.0 (19.5) | -46.0 (21.4)
  Change at Week 36: number analyzed (Participants) | 347 | 177 | 178 | 324
  Change at Week 36 | -53.0 (20.5) | -51.0 (22.3) | -52.0 (18.6) | -51.0 (20.6)
  Change at Week 52: number analyzed (Participants) | 332 | 169 | 171 | 307
  Change at Week 52 | -56.0 (20.0) | -54.0 (20.7) | -55.0 (17.5) | -51.0 (20.2)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-12.0 to -6.0], Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-9.0 to -2.0], Standard Error of Mean 1.6
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.0, 95% CI 2-sided [-11.0 to -5.0], Standard Error of Mean 1.6
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -11.0, 95% CI 2-sided [-13.0 to -8.0], Standard Error of Mean 1.4
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.0, 95% CI 2-sided [-11.0 to -4.0], Standard Error of Mean 1.7
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.0, 95% CI 2-sided [-11.0 to -5.0], Standard Error of Mean 1.7
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-12.0 to -7.0], Standard Error of Mean 1.3
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-9.0 to -2.0], Standard Error of Mean 1.6
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-8.0 to -2.0], Standard Error of Mean 1.6
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-8.0 to -3.0], Standard Error of Mean 1.2
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.007, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-7.0 to -1.0], Standard Error of Mean 1.5
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.046, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-6.0 to -0.0], Standard Error of Mean 1.5
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-6.0 to -1.0], Standard Error of Mean 1.2
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.44, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-4.0 to 2.0], Standard Error of Mean 1.4
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.21, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-5.0 to 1.0], Standard Error of Mean 1.4
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-7.0 to -3.0], Standard Error of Mean 1.1
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.029, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-6.0 to -0.0], Standard Error of Mean 1.4
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.010, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-6.0 to -1.0], Standard Error of Mean 1.4

16. Secondary Outcome: Change From Baseline in Individual ACR Component: Subject's Pain Assessment at Weeks 2, 4, 12, 24, 36, and 52
Description: The participant assessed their pain severity using a VAS on a scale of 0 ( no pain) to 100 (severe pain). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 414 | 207 | 210 | 416
  Baseline | 64.0 (22.0) | 67.0 (22.1) | 67.0 (18.4) | 66.0 (21.4)
  Change at Week 2: number analyzed (Participants) | 400 | 202 | 202 | 405
  Change at Week 2 | -18.0 (22.2) | -15.0 (20.3) | -17.0 (21.6) | -7.0 (20.1)
  Change at Week 4: number analyzed (Participants) | 405 | 200 | 205 | 403
  Change at Week 4 | -26.0 (24.8) | -22.0 (23.7) | -24.0 (25.3) | -14.0 (23.6)
  Change at Week 12: number analyzed (Participants) | 389 | 197 | 193 | 389
  Change at Week 12 | -37.0 (27.1) | -31.0 (26.9) | -32.0 (28.3) | -26.0 (27.0)
  Change at Week 24: number analyzed (Participants) | 372 | 190 | 185 | 370
  Change at Week 24 | -41.0 (28.0) | -37.0 (27.8) | -39.0 (26.1) | -34.0 (27.6)
  Change at Week 36: number analyzed (Participants) | 348 | 178 | 179 | 326
  Change at Week 36 | -43.0 (28.0) | -40.0 (28.8) | -38.0 (25.6) | -38.0 (29.3)
  Change at Week 52: number analyzed (Participants) | 332 | 169 | 171 | 307
  Change at Week 52 | -45.0 (27.9) | -43.0 (27.9) | -44.0 (24.2) | -37.0 (30.5)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -12.0, 95% CI 2-sided [-15.0 to -9.0], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.0, 95% CI 2-sided [-11.0 to -5.0], Standard Error of Mean 1.7
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-13.0 to -6.0], Standard Error of Mean 1.7
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -13.0, 95% CI 2-sided [-16.0 to -10.0], Standard Error of Mean 1.5
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-11.0 to -4.0], Standard Error of Mean 1.9
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-13.0 to -6.0], Standard Error of Mean 1.9
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -12.0, 95% CI 2-sided [-15.0 to -8.0], Standard Error of Mean 1.7
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p = 0.019, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5, 95.0% CI 2-sided [-9.0 to -1.0], Standard Error of Mean 2.1
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.007, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-10.0 to -2.0], Standard Error of Mean 2.1
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-12.0 to -5.0], Standard Error of Mean 1.7
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.13, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-7.0 to 1.0], Standard Error of Mean 2.0
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.047, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-8.0 to -0.0], Standard Error of Mean 2.0
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-11.0 to -4.0], Standard Error of Mean 1.8
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.34, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-6.0 to 2.0], Standard Error of Mean 2.1
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.46, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-6.0 to 3.0], Standard Error of Mean 2.1
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.0, 95% CI 2-sided [-12.0 to -5.0], Standard Error of Mean 1.8
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.030, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-9.0 to -0.0], Standard Error of Mean 2.2
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-12.0 to -3.0], Standard Error of Mean 2.2

17. Secondary Outcome: Change From Baseline in Individual ACR Component: High-Sensitivity C-Reactive Protein (hsCRP) at Weeks 2, 4, 12, 24, 36, and 52
Time Frame: Baseline; Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
mg/L
  Baseline | 18.04 (25.289) | 17.72 (27.419) | 17.32 (23.228) | 16.86 (24.353)
  Change at Week 2: number analyzed (Participants) | 404 | 200 | 204 | 400
  Change at Week 2 | -12.89 (23.401) | -9.40 (18.930) | -10.97 (20.249) | -0.99 (14.392)
  Change at Week 4: number analyzed (Participants) | 404 | 200 | 203 | 402
  Change at Week 4 | -13.79 (23.569) | -11.53 (20.596) | -10.95 (23.319) | -3.18 (18.534)
  Change at Week 12: number analyzed (Participants) | 388 | 196 | 190 | 383
  Change at Week 12 | -13.77 (23.585) | -11.02 (20.272) | -12.04 (24.690) | -7.23 (21.823)
  Change at Week 24: number analyzed (Participants) | 374 | 190 | 186 | 368
  Change at Week 24 | -13.43 (27.086) | -10.85 (24.458) | -12.66 (24.525) | -7.47 (23.511)
  Change at Week 36: number analyzed (Participants) | 348 | 177 | 177 | 321
  Change at Week 36 | -12.99 (26.823) | -12.64 (22.736) | -11.52 (26.863) | -8.74 (23.579)
  Change at Week 52: number analyzed (Participants) | 332 | 170 | 170 | 307
  Change at Week 52 | -13.84 (25.180) | -11.61 (23.857) | -12.29 (23.090) | -7.96 (23.835)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -10.78, 95% CI 2-sided [-12.71 to -8.85], Standard Error of Mean 0.983
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.76, 95% CI 2-sided [-11.13 to -6.39], Standard Error of Mean 1.207
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.64, 95% CI 2-sided [-12.00 to -7.29], Standard Error of Mean 1.200
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.92, 95% CI 2-sided [-11.65 to -8.19], Standard Error of Mean 0.884
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.34, 95% CI 2-sided [-10.47 to -6.21], Standard Error of Mean 1.086
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.33, 95% CI 2-sided [-9.45 to -5.21], Standard Error of Mean 1.080
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.98, 95% CI 2-sided [-7.56 to -4.39], Standard Error of Mean 0.808
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.21, 95% CI 2-sided [-6.14 to -2.27], Standard Error of Mean 0.987
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.34, 95% CI 2-sided [-6.29 to -2.39], Standard Error of Mean 0.993
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.27, 95% CI 2-sided [-7.24 to -3.31], Standard Error of Mean 1.003
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.007, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.29, 95% CI 2-sided [-5.68 to -0.89], Standard Error of Mean 1.222
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.61, 95% CI 2-sided [-7.02 to -2.20], Standard Error of Mean 1.229
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.44, 95% CI 2-sided [-5.35 to -1.53], Standard Error of Mean 0.974
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.004, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.40, 95% CI 2-sided [-5.72 to -1.09], Standard Error of Mean 1.180
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.072, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.12, 95% CI 2-sided [-4.44 to 0.19], Standard Error of Mean 1.180
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.79, 95% CI 2-sided [-6.34 to -3.24], Standard Error of Mean 0.789
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.01, 95% CI 2-sided [-4.88 to -1.13], Standard Error of Mean 0.957
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.77, 95% CI 2-sided [-5.65 to -1.89], Standard Error of Mean 0.957

18. Secondary Outcome: Percentage of Participants Who Achieved an Improvement (Decrease) in the HAQ-DI Score ≥ 0.22 at Weeks 2, 4, 12, 24, 36, and 52
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0-3 [0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0-3 [0 (no disability) to 3 (completely disabled)] when 6 or more categories are non-missing, so total possible score is 3. Improvement is defined as reduction in HAQ-DI, (baseline value - postbaseline value) ≥ 0.22. If more than 2 categories are missing, the HAQ-DI score is set to missing. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of participants
  Week 2: number analyzed (Participants) | 402 | 200 | 204 | 410
  Week 2 | 61.9 [57.1 to 66.8] | 58.5 [51.4 to 65.6] | 53.9 [46.8 to 61.0] | 42.2 [37.3 to 47.1]
  Week 4: number analyzed (Participants) | 402 | 200 | 204 | 410
  Week 4 | 72.4 [67.9 to 76.9] | 61.0 [54.0 to 68.0] | 68.6 [62.0 to 75.2] | 53.9 [49.0 to 58.8]
  Week 12: number analyzed (Participants) | 402 | 200 | 204 | 410
  Week 12 | 80.3 [76.3 to 84.4] | 74.5 [68.2 to 80.8] | 74.0 [67.8 to 80.3] | 69.8 [65.2 to 74.3]
  Week 24: number analyzed (Participants) | 402 | 200 | 204 | 410
  Week 24 | 76.6 [72.4 to 80.9] | 78.5 [72.6 to 84.4] | 77.0 [70.9 to 83.0] | 73.9 [69.5 to 78.3]
  Week 36: number analyzed (Participants) | 402 | 200 | 204 | 410
  Week 36 | 73.4 [68.9 to 77.8] | 76.5 [70.4 to 82.6] | 73.5 [67.2 to 79.8] | 67.1 [62.4 to 71.7]
  Week 52: number analyzed (Participants) | 402 | 200 | 204 | 410
  Week 52 | 70.9 [66.3 to 75.5] | 71.5 [65.0 to 78.0] | 70.6 [64.1 to 77.1] | 61.0 [56.1 to 65.8]
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.7, 95% CI 2-sided [12.8 to 26.7]
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.3, 95% CI 2-sided [7.6 to 25.0]
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 2; Test type: Superiority; p = 0.004, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.7, 95% CI 2-sided [3.0 to 20.4]
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.5, 95% CI 2-sided [11.7 to 25.2]
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p = 0.083, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.1, 95% CI 2-sided [-1.6 to 15.8]
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.7, 95% CI 2-sided [6.4 to 23.1]
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 10.6, 95% CI 2-sided [4.4 to 16.7]
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p = 0.22, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 4.7, 95% CI 2-sided [-3.1 to 12.6]
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 12; Test type: Superiority; p = 0.25, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 4.3, 95% CI 2-sided [-3.6 to 12.1]
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p = 0.35, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 2.7, 95% CI 2-sided [-3.5 to 8.9]
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p = 0.20, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 4.6, 95% CI 2-sided [-2.9 to 12.1]
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24; Test type: Superiority; p = 0.36, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 3.1, 95% CI 2-sided [-4.5 to 10.6]
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.043, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 6.3, 95% CI 2-sided [-0.2 to 12.8]
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.015, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 9.4, 95% CI 2-sided [1.6 to 17.2]
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.085, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 6.5, 95% CI 2-sided [-1.5 to 14.4]
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p = 0.002, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 9.9, 95% CI 2-sided [3.2 to 16.6]
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p = 0.010, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 10.5, 95% CI 2-sided [2.3 to 18.7]
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52; Test type: Superiority; p = 0.014, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 9.6, 95% CI 2-sided [1.4 to 17.8]

19. Secondary Outcome: Change From Baseline in DAS28 (CRP) at Weeks 2, 4, 12, 24, 36, and 52
Description: The DAS28 score is a measure of the participant's disease activity calculated using the TJC (28 joints), SJC (28 joints), Patient's Global Assessment of Disease Activity (VAS: 0 = no disease activity to 100 = maximum disease activity), and CRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline | 5.7 (0.99) | 5.7 (1.04) | 5.8 (0.94) | 5.7 (1.00)
  Change at Week 2: number analyzed (Participants) | 399 | 199 | 200 | 396
  Change at Week 2 | -1.3 (1.06) | -1.1 (0.92) | -1.4 (1.12) | -0.6 (0.87)
  Change at Week 4: number analyzed (Participants) | 403 | 199 | 202 | 401
  Change at Week 4 | -1.9 (1.26) | -1.6 (1.14) | -1.8 (1.20) | -1.0 (1.04)
  Change at Week 12: number analyzed (Participants) | 386 | 195 | 189 | 380
  Change at Week 12 | -2.7 (1.31) | -2.5 (1.28) | -2.6 (1.26) | -1.9 (1.21)
  Change at Week 24: number analyzed (Participants) | 374 | 190 | 183 | 368
  Change at Week 24 | -3.2 (1.31) | -2.9 (1.30) | -3.0 (1.16) | -2.5 (1.29)
  Change at Week 36: number analyzed (Participants) | 347 | 177 | 177 | 321
  Change at Week 36 | -3.3 (1.28) | -3.0 (1.26) | -3.2 (1.12) | -2.9 (1.22)
  Change at Week 52: number analyzed (Participants) | 332 | 170 | 169 | 307
  Change at Week 52 | -3.4 (1.23) | -3.1 (1.24) | -3.3 (1.11) | -2.8 (1.29)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-0.9 to -0.6], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.4], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-0.9 to -0.6], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-1.1 to -0.8], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-0.9 to -0.5], Standard Error of Mean 0.09
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-1.0 to -0.7], Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-1.0 to -0.7], Standard Error of Mean 0.08
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-0.8 to -0.4], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-0.9 to -0.5], Standard Error of Mean 0.10
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-0.9 to -0.6], Standard Error of Mean 0.08
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.3], Standard Error of Mean 0.10
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.3], Standard Error of Mean 0.10
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.6 to -0.3], Standard Error of Mean 0.08
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.033, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.4 to -0.0], Standard Error of Mean 0.10
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.2], Standard Error of Mean 0.10
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-0.8 to -0.5], Standard Error of Mean 0.08
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.6 to -0.2], Standard Error of Mean 0.10
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.7 to -0.3], Standard Error of Mean 0.10

20. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) ≤ 3.2 at Weeks 4, 12, 24, and 52
Description: as for outcome 3
Time Frame: Weeks 4, 12, 24, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of participants
  Week 4 | 30.8 [26.2 to 35.3] | 23.7 [17.6 to 29.7] | 31.9 [25.4 to 38.4] | 12.0 [8.8 to 15.3]
  Week 12 | 55.8 [50.9 to 60.7] | 50.2 [43.2 to 57.3] | 48.1 [41.1 to 55.1] | 28.6 [24.1 to 33.1]
  Week 24 | 68.8 [64.2 to 73.3] | 62.8 [56.0 to 69.6] | 60.0 [53.1 to 66.9] | 46.2 [41.2 to 51.1]
  Week 52 | 69.0 [64.4 to 73.6] | 59.9 [53.0 to 66.8] | 65.7 [59.1 to 72.4] | 47.6 [42.7 to 52.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.8, 95% CI 2-sided [13.1 to 24.4]
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.7, 95% CI 2-sided [4.7 to 18.6]
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.9, 95% CI 2-sided [12.5 to 27.3]
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 27.2, 95% CI 2-sided [20.5 to 33.9]
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 21.6, 95% CI 2-sided [13.2 to 30.1]
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 19.5, 95% CI 2-sided [11.1 to 27.9]
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 22.6, 95% CI 2-sided [15.8 to 29.4]
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.6, 95% CI 2-sided [8.1 to 25.2]
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 13.8, 95% CI 2-sided [5.3 to 22.4]
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 21.4, 95% CI 2-sided [14.6 to 28.2]
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p = 0.003, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.3, 95% CI 2-sided [3.7 to 20.9]
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.1, 95% CI 2-sided [9.7 to 26.5]

21. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) < 2.6 at Weeks 2, 4, 12, 36, and 52
Description: as for outcome 3
Time Frame: Weeks 2, 4, 12, 36, and 52
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of participants
  Week 2 | 7.2 [4.6 to 9.8] | 4.3 [1.3 to 7.4] | 10.0 [5.7 to 14.3] | 1.0 [0.0 to 2.0]
  Week 4 | 16.6 [12.9 to 20.3] | 15.0 [9.9 to 20.1] | 19.5 [13.9 to 25.1] | 4.8 [2.6 to 7.0]
  Week 12 | 39.7 [34.8 to 44.5] | 31.9 [25.3 to 38.5] | 29.5 [23.1 to 35.9] | 17.1 [13.3 to 20.8]
  Week 36 | 52.6 [47.7 to 57.6] | 42.0 [35.1 to 49.0] | 43.3 [36.4 to 50.3] | 34.4 [29.7 to 39.1]
  Week 52 | 53.4 [48.5 to 58.3] | 43.0 [36.0 to 50.0] | 46.2 [39.2 to 53.2] | 31.5 [26.9 to 36.1]
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 6.3, 95% CI 2-sided [3.4 to 9.1]
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 2; Test type: Superiority; p = 0.010, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 3.4, 95% CI 2-sided [0.1 to 6.7]
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 2; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 9.0, 95% CI 2-sided [4.5 to 13.6]
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.8, 95% CI 2-sided [7.4 to 16.1]
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 10.2, 95% CI 2-sided [4.5 to 15.8]
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.7, 95% CI 2-sided [8.6 to 20.8]
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 22.6, 95% CI 2-sided [16.4 to 28.8]
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.8, 95% CI 2-sided [7.1 to 22.5]
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.5, 95% CI 2-sided [4.9 to 20.0]
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.3, 95% CI 2-sided [11.4 to 25.1]
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.056, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.7, 95% CI 2-sided [-0.8 to 16.1]
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 36; Test type: Superiority; p = 0.023, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 9.0, 95% CI 2-sided [0.5 to 17.4]
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 21.9, 95% CI 2-sided [15.1 to 28.7]
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52; Test type: Superiority; p = 0.004, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 11.5, 95% CI 2-sided [3.1 to 20.0]
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.7, 95% CI 2-sided [6.3 to 23.1]

22. Secondary Outcome: ACR N Percent Improvement (ACR-N) Response at Weeks 2, 4, 12, 24, 36, and 52
Description: ACR-N is defined as the smallest percentage improvement from baseline in swollen joints, tender joints and the median of the following 5 items (PGA, SGA, subject's pain assessment, HAQ-DI and CRP). It has a range between 0 and 100%. PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions,8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]. If this calculation results in a negative value, then the ACR-N is set to 0. The ACR-N value indicates an improvement of N%, with higher numbers indicating greater improvement.
Time Frame: Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percent improvement
  Week 2: number analyzed (Participants) | 386 | 191 | 197 | 387
  Week 2 | 20.8 (21.42) | 17.8 (20.07) | 20.9 (23.19) | 8.9 (14.95)
  Week 4: number analyzed (Participants) | 389 | 192 | 193 | 395
  Week 4 | 34.1 (27.78) | 27.6 (24.81) | 29.4 (27.86) | 17.2 (21.43)
  Week 12: number analyzed (Participants) | 377 | 188 | 185 | 375
  Week 12 | 52.6 (29.91) | 46.1 (31.46) | 48.6 (30.50) | 34.3 (28.07)
  Week 24: number analyzed (Participants) | 365 | 181 | 180 | 359
  Week 24 | 62.8 (28.40) | 58.1 (30.19) | 59.7 (29.35) | 49.0 (29.46)
  Week 36: number analyzed (Participants) | 341 | 170 | 173 | 315
  Week 36 | 65.8 (28.50) | 58.7 (30.99) | 62.1 (28.12) | 57.3 (29.16)
  Week 52: number analyzed (Participants) | 327 | 163 | 166 | 304
  Week 52 | 69.6 (27.38) | 63.6 (29.19) | 67.4 (26.60) | 57.1 (29.59)

23. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response at Weeks 2, 4, 12, 24, 36, and 52
Description: Good Response: DAS28(CRP) at visit ≤3.2 and improvement from baseline >1.2. Moderate Response: DAS28(CRP) at visit ≤3.2 and improvement from baseline >0.6 and ≤1.2; DAS28(CRP) at visit >3.2 and ≤5.1 and improvement from baseline >0.6; DAS 28(CRP) at visit >5.1 and improvement from baseline >1.2.
  No Response: DAS28(CRP) at visit ≤5.1 and improvement from baseline ≤0.6; DAS 28(CRP) >5.1 at visit and improvement from baseline ≤1.2.
Time Frame: Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
Participants
  Week 2: number analyzed (Participants) | 399 | 199 | 200 | 396
  Week 2: Good Response | 66 | 21 | 35 | 20
  Week 2: Moderate Response | 199 | 92 | 88 | 118
  Week 2: No Response | 134 | 86 | 77 | 258
  Week 4: number analyzed (Participants) | 403 | 199 | 202 | 401
  Week 4: Good Response | 120 | 45 | 63 | 45
  Week 4: Moderate Response | 206 | 104 | 97 | 161
  Week 4: No Response | 77 | 50 | 42 | 195
  Week 12: number analyzed (Participants) | 386 | 195 | 189 | 380
  Week 12: Good Response | 230 | 100 | 98 | 116
  Week 12: Moderate Response | 130 | 79 | 77 | 190
  Week 12: No Response | 26 | 16 | 14 | 74
  Week 24: number analyzed (Participants) | 374 | 190 | 183 | 368
  Week 24: Good Response | 283 | 127 | 126 | 186
  Week 24: Moderate Response | 82 | 55 | 52 | 153
  Week 24: No Response | 9 | 8 | 5 | 29
  Week 36: number analyzed (Participants) | 347 | 177 | 177 | 321
  Week 36: Good Response | 276 | 118 | 124 | 208
  Week 36: Moderate Response | 64 | 54 | 51 | 106
  Week 36: No Response | 7 | 5 | 2 | 7
  Week 52: number analyzed (Participants) | 332 | 170 | 169 | 307
  Week 52: Good Response | 286 | 123 | 136 | 194
  Week 52: Moderate Response | 43 | 43 | 30 | 102
  Week 52: No Response | 3 | 4 | 3 | 11

24. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 2, 4, 12, 24, 36, and 52
Description: CDAI is calculated using formula: CDAI = TJC28 + SJC28 + SGA + PGA. PGA and SGA are assessed using a VAS on a scale of 0-10 [0 and 10 indicating no disease activity and maximum disease activity]. CDAI can range from 0 to 76, with higher score indicating more severe disease activity status.
Time Frame: Baseline; Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline | 39.5 (12.77) | 39.2 (12.69) | 40.0 (12.63) | 40.2 (12.50)
  Change at Week 2: number analyzed (Participants) | 396 | 199 | 201 | 401
  Change at Week 2 | -13.6 (12.05) | -12.0 (10.54) | -13.9 (12.53) | -8.5 (11.33)
  Change at Week 4: number analyzed (Participants) | 401 | 200 | 198 | 402
  Change at Week 4 | -19.9 (13.64) | -17.8 (12.06) | -18.4 (12.96) | -13.3 (12.61)
  Change at Week 12: number analyzed (Participants) | 388 | 195 | 191 | 384
  Change at Week 12 | -27.8 (13.60) | -26.1 (13.00) | -27.5 (13.55) | -22.7 (13.38)
  Change at Week 24: number analyzed (Participants) | 372 | 187 | 184 | 364
  Change at Week 24 | -31.3 (13.19) | -30.0 (13.32) | -31.3 (12.57) | -28.2 (13.43)
  Change at Week 36: number analyzed (Participants) | 347 | 177 | 178 | 324
  Change at Week 36 | -32.2 (13.37) | -30.8 (12.84) | -32.7 (12.16) | -31.3 (12.66)
  Change at Week 52: number analyzed (Participants) | 332 | 169 | 171 | 307
  Change at Week 52 | -33.8 (13.00) | -31.9 (12.22) | -33.6 (12.28) | -31.2 (13.12)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.7, 95% CI 2-sided [-7.3 to -4.1], Standard Error of Mean 0.82
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.4, 95% CI 2-sided [-6.4 to -2.4], Standard Error of Mean 1.01
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.7, 95% CI 2-sided [-7.7 to -3.7], Standard Error of Mean 1.01
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.3, 95% CI 2-sided [-8.9 to -5.6], Standard Error of Mean 0.83
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.3, 95% CI 2-sided [-7.3 to -3.3], Standard Error of Mean 1.02
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.7, 95% CI 2-sided [-7.8 to -3.7], Standard Error of Mean 1.02
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.8, 95% CI 2-sided [-7.3 to -4.4], Standard Error of Mean 0.72
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.4, 95% CI 2-sided [-6.1 to -2.7], Standard Error of Mean 0.88
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.1, 95% CI 2-sided [-6.8 to -3.4], Standard Error of Mean 0.88
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.1, 95% CI 2-sided [-5.3 to -2.9], Standard Error of Mean 0.61
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.8, 95% CI 2-sided [-4.3 to -1.3], Standard Error of Mean 0.75
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.9, 95% CI 2-sided [-4.4 to -1.4], Standard Error of Mean 0.75
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.2, 95% CI 2-sided [-3.4 to -1.1], Standard Error of Mean 0.59
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.36, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.65, 95% CI 2-sided [-2.0 to 0.8], Standard Error of Mean 0.71
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.009, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.9, 95% CI 2-sided [-3.3 to -0.5], Standard Error of Mean 0.72
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.3, 95% CI 2-sided [-4.5 to -2.2], Standard Error of Mean 0.56
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.042, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.4, 95% CI 2-sided [-2.7 to -0.1], Standard Error of Mean 0.69
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.4, 95% CI 2-sided [-3.7 to -1.0], Standard Error of Mean 0.69

25. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 2, 4, 12, 24, 36, and 52
Description: SDAI is a composite measure that sums the TJC28, SJC28, SGA, PGA, and the hsCRP (in mg/dL). PGA and SGA assessed using VAS on a scale of 0-10 [0 and 10 indicating no disease activity and maximum disease activity]. Higher score indicates more severe disease activity status and total possible score is 86. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline | 41.3 (13.41) | 41.0 (13.53) | 41.8 (13.09) | 41.9 (13.39)
  Change at Week 2: number analyzed (Participants) | 394 | 197 | 200 | 392
  Change at Week 2 | -14.9 (12.45) | -12.9 (10.84) | -15.0 (12.82) | -8.6 (11.49)
  Change at Week 4: number analyzed (Participants) | 397 | 199 | 196 | 399
  Change at Week 4 | -21.3 (14.17) | -19.0 (12.58) | -19.6 (13.38) | -13.7 (12.83)
  Change at Week 12: number analyzed (Participants) | 384 | 194 | 188 | 378
  Change at Week 12 | -29.2 (14.05) | -27.1 (13.59) | -28.6 (14.02) | -23.5 (13.82)
  Change at Week 24: number analyzed (Participants) | 372 | 187 | 183 | 362
  Change at Week 24 | -32.7 (13.83) | -31.1 (14.09) | -32.7 (13.14) | -29.0 (14.09)
  Change at Week 36: number analyzed (Participants) | 346 | 176 | 176 | 318
  Change at Week 36 | -33.5 (14.02) | -32.1 (13.61) | -33.9 (12.67) | -32.3 (13.47)
  Change at Week 52: number analyzed (Participants) | 332 | 169 | 169 | 307
  Change at Week 52 | -35.2 (13.68) | -33.0 (13.12) | -35.0 (12.69) | -32.0 (14.14)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.8, 95% CI 2-sided [-8.5 to -5.2], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.3, 95% CI 2-sided [-7.3 to -3.3], Standard Error of Mean 1.04
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.7, 95% CI 2-sided [-8.8 to -4.7], Standard Error of Mean 1.03
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.3, 95% CI 2-sided [-9.9 to -6.6], Standard Error of Mean 0.85
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.2, 95% CI 2-sided [-8.2 to -4.1], Standard Error of Mean 1.04
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.5, 95% CI 2-sided [-8.5 to -4.5], Standard Error of Mean 1.04
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.5, 95% CI 2-sided [-8.0 to -5.1], Standard Error of Mean 0.74
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.8, 95% CI 2-sided [-6.5 to -3.0], Standard Error of Mean 0.90
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.6, 95% CI 2-sided [-7.4 to -3.8], Standard Error of Mean 0.90
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.6, 95% CI 2-sided [-5.9 to -3.4], Standard Error of Mean 0.64
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.1, 95% CI 2-sided [-4.6 to -1.6], Standard Error of Mean 0.78
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.4, 95% CI 2-sided [-4.9 to -1.9], Standard Error of Mean 0.79
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.6, 95% CI 2-sided [-3.8 to -1.4], Standard Error of Mean 0.61
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.23, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-2.4 to 0.6], Standard Error of Mean 0.74
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.005, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.1, 95% CI 2-sided [-3.6 to -0.6], Standard Error of Mean 0.75
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.8, 95% CI 2-sided [-5.0 to -2.6], Standard Error of Mean 0.60
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.021, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.7, 95% CI 2-sided [-3.1 to -0.3], Standard Error of Mean 0.73
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.8, 95% CI 2-sided [-4.3 to -1.4], Standard Error of Mean 0.73

26. Secondary Outcome: Percentage of Participants With no Radiographic Progression From Baseline at Weeks 24, and 52
Description: Participant's radiographs of bilateral hands, wrists and feet are taken and evaluated through central review using the mTSS method. No radiographic progression is defined by the change from baseline in mTSS and is reported for the following categories: Change in mTSS ≤ 0.5, Change in mTSS ≤ 0 and Change in mTSS ≤ smallest detectable change (SDC).
Time Frame: Baseline; Weeks 24, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of participants
  Week 24: Change in mTSS ≤ 0.5: number analyzed (Participants) | 355 | 184 | 173 | 356
  Week 24: Change in mTSS ≤ 0.5 | 89.6 [86.3 to 92.9] | 87.0 [81.8 to 92.1] | 89.6 [84.8 to 94.4] | 82.0 [77.9 to 86.2]
  Week 24: Change in mTSS ≤ 0: number analyzed (Participants) | 355 | 184 | 173 | 356
  Week 24: Change in mTSS ≤ 0 | 80.6 [76.3 to 84.8] | 76.6 [70.2 to 83.0] | 82.7 [76.7 to 88.6] | 72.5 [67.7 to 77.3]
  Week 24: Change in mTSS ≤ SDC (1.53): number analyzed (Participants) | 355 | 184 | 173 | 356
  Week 24: Change in mTSS ≤ SDC (1.53) | 95.2 [92.8 to 97.6] | 93.5 [89.6 to 97.3] | 96.0 [92.7 to 99.2] | 91.6 [88.5 to 94.6]
  Week 52: Change in mTSS ≤ 0.5: number analyzed (Participants) | 345 | 176 | 166 | 330
  Week 52: Change in mTSS ≤ 0.5 | 88.1 [84.6 to 91.7] | 85.8 [80.4 to 91.2] | 84.3 [78.5 to 90.2] | 77.9 [73.2 to 82.5]
  Week 52: Change in mTSS ≤ 0: number analyzed (Participants) | 345 | 176 | 166 | 330
  Week 52: Change in mTSS ≤ 0 | 80.6 [76.3 to 84.9] | 76.1 [69.6 to 82.7] | 77.1 [70.4 to 83.8] | 70.6 [65.5 to 75.7]
  Week 52: Change in mTSS ≤ SDC (1.77): number analyzed (Participants) | 345 | 176 | 166 | 330
  Week 52: Change in mTSS ≤ SDC (1.77) | 94.2 [91.6 to 96.8] | 94.9 [91.3 to 98.4] | 89.2 [84.1 to 94.2] | 86.7 [82.8 to 90.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24 for Change in mTSS <= 0.5; Test type: Superiority; p = 0.006, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, and stratification factors in the model; Difference in Response Rates = 7.6, 95% CI 2-sided [2.2 to 12.9]
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24 for Change in mTSS <= 0.5; Test type: Superiority; p = 0.16, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, and stratification factors in the model; Difference in Response Rates = 4.9, 95% CI 2-sided [-1.8 to 11.6]
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24 for Change in mTSS <= 0.5; Test type: Superiority; p = 0.029, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, and stratification factors in the model; Difference in Response Rates = 7.6, 95% CI 2-sided [1.1 to 14.1]
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24 for Change in mTSS <= 0; Test type: Superiority; p = 0.015, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, and stratification factors in the model; Difference in Response Rates = 8.1, 95% CI 2-sided [1.6 to 14.6]
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24 for Change in mTSS <= 0; Test type: Superiority; p = 0.33, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, and stratification factors in the model; Difference in Response Rates = 4.2, 95% CI 2-sided [-3.9 to 12.2]
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24 for Change in mTSS <= 0; Test type: Superiority; p = 0.013, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, and stratification factors in the model; Difference in Response Rates = 10.2, 95% CI 2-sided [2.5 to 17.9]
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 24 for Change in mTSS <= SDC (1.53); Test type: Superiority; p = 0.074, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, and stratification factors in the model; Difference in Response Rates = 3.6, 95% CI 2-sided [-0.3 to 7.6]
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 24 for Change in mTSS <= SDC (1.53); Test type: Superiority; p = 0.49, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, and stratification factors in the model; Difference in Response Rates = 1.9, 95% CI 2-sided [-3.1 to 6.9]
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 24 for Change in mTSS <= SDC (1.53); Test type: Superiority; p = 0.075, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, and stratification factors in the model; Difference in Response Rates = 4.4, 95% CI 2-sided [-0.2 to 8.9]
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52 for Change in mTSS <= 0.5; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups, stratification factors and campaign groups in the model; Difference in Response Rates = 10.2, 95% CI 2-sided [4.3 to 16.2]
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52 for Change in mTSS <= 0.5; Test type: Superiority; p = 0.045, Regression, Logistic — [p-value comment as in outcome 26, analysis 10]; Difference in Response Rates = 7.9, 95% CI 2-sided [0.7 to 15.2]
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52 for Change in mTSS <= 0.5; Test type: Superiority; p = 0.100, Regression, Logistic — [p-value comment as in outcome 26, analysis 10]; Difference in Response Rates = 6.5, 95% CI 2-sided [-1.1 to 14.0]
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52 for Change in mTSS <= 0; Test type: Superiority; p = 0.004, Regression, Logistic — [p-value comment as in outcome 26, analysis 10]; Difference in Response Rates = 10.0, 95% CI 2-sided [3.2 to 16.7]
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52 for Change in mTSS <= 0; Test type: Superiority; p = 0.25, Regression, Logistic — [p-value comment as in outcome 26, analysis 10]; Difference in Response Rates = 5.5, 95% CI 2-sided [-2.9 to 14.0]
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52 for Change in mTSS <= 0; Test type: Superiority; p = 0.14, Regression, Logistic — [p-value comment as in outcome 26, analysis 10]; Difference in Response Rates = 6.5, 95% CI 2-sided [-2.0 to 15.0]
Statistical Analysis 16: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; Filgotinib 200 mg + MTX vs MTX Monotherapy at Week 52 for Change in mTSS <= SDC (1.77); Test type: Superiority; p = 0.002, Regression, Logistic — [p-value comment as in outcome 26, analysis 10]; Difference in Response Rates = 7.5, 95% CI 2-sided [2.8 to 12.3]
Statistical Analysis 17: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; Filgotinib 100 mg + MTX vs MTX Monotherapy at Week 52 for Change in mTSS <= SDC (1.77); Test type: Superiority; p = 0.008, Regression, Logistic — [p-value comment as in outcome 26, analysis 10]; Difference in Response Rates = 8.2, 95% CI 2-sided [2.9 to 13.6]
Statistical Analysis 18: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; Filgotinib 200 mg Monotherapy vs MTX Monotherapy at Week 52 for Change in mTSS <= SDC (1.77); Test type: Superiority; p = 0.47, Regression, Logistic — [p-value comment as in outcome 26, analysis 10]; Difference in Response Rates = 2.5, 95% CI 2-sided [-3.9 to 8.9]

27. Secondary Outcome: SF-36 PCS Score at Weeks 4, 12, 24, 36, and 52
Description: The SF-36 is a 36-item, self-reported, generic, comprehensive, and health-related quality of life questionnaire based on 8 health domains in 2 components: physical well-being (physical functioning, role-physical, bodily pain, general health perceptions), mental well-being (vitality, social functioning, role-emotional, and mental health). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with highest possible score of 100. Higher scores indicate better health status or functioning.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Week 4: number analyzed (Participants) | 408 | 203 | 205 | 411
  Week 4 | 40.6 (8.04) | 39.2 (8.86) | 39.6 (8.46) | 37.0 (8.13)
  Week 12: number analyzed (Participants) | 394 | 198 | 195 | 389
  Week 12 | 45.0 (8.42) | 42.9 (9.71) | 42.7 (9.90) | 40.9 (8.10)
  Week 24: number analyzed (Participants) | 375 | 190 | 187 | 371
  Week 24 | 46.3 (8.16) | 44.8 (9.39) | 44.1 (9.42) | 43.0 (8.36)
  Week 36: number analyzed (Participants) | 348 | 178 | 179 | 327
  Week 36 | 46.6 (8.17) | 45.2 (9.42) | 45.0 (8.89) | 44.4 (8.39)
  Week 52: number analyzed (Participants) | 333 | 169 | 172 | 307
  Week 52 | 47.4 (8.35) | 45.6 (9.02) | 45.9 (9.40) | 44.5 (8.32)

28. Secondary Outcome: Change From Baseline in SF-36 PCS Score at Weeks 4, 12, 36, and 52
Description: as for outcome 5
Time Frame: Baseline; Weeks 4, 12, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 414 | 207 | 208 | 416
  Baseline | 33.9 (7.48) | 33.7 (8.00) | 33.6 (7.70) | 33.3 (7.28)
  Change at Week 4: number analyzed (Participants) | 406 | 203 | 203 | 411
  Change at Week 4 | 6.8 (6.86) | 5.3 (6.90) | 5.9 (7.53) | 3.8 (6.38)
  Change at Week 12: number analyzed (Participants) | 392 | 198 | 193 | 389
  Change at Week 12 | 11.2 (8.66) | 9.1 (8.82) | 8.9 (9.17) | 7.6 (7.64)
  Change at Week 36: number analyzed (Participants) | 346 | 178 | 177 | 327
  Change at Week 36 | 12.4 (9.30) | 11.7 (8.52) | 11.2 (8.54) | 11.3 (9.04)
  Change at Week 52: number analyzed (Participants) | 331 | 169 | 170 | 307
  Change at Week 52 | 13.4 (9.62) | 12.0 (8.47) | 11.9 (9.22) | 11.2 (9.49)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.2, 95% CI 2-sided [2.4 to 4.1], Standard Error of Mean 0.45
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.8, 95% CI 2-sided [0.7 to 2.8], Standard Error of Mean 0.55
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.3, 95% CI 2-sided [1.3 to 3.4], Standard Error of Mean 0.55
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.7, 95% CI 2-sided [2.7 to 4.8], Standard Error of Mean 0.54
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p = 0.008, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.7, 95% CI 2-sided [0.5 to 3.0], Standard Error of Mean 0.66
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.023, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.5, 95% CI 2-sided [0.2 to 2.8], Standard Error of Mean 0.66
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.8, 95% CI 2-sided [0.6 to 2.9], Standard Error of Mean 0.59
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.38, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.6, 95% CI 2-sided [-0.8 to 2.0], Standard Error of Mean 0.71
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.59, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.4, 95% CI 2-sided [-1.0 to 1.8], Standard Error of Mean 0.72
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.8, 95% CI 2-sided [1.6 to 4.0], Standard Error of Mean 0.62
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.11, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.2, 95% CI 2-sided [-0.3 to 2.7], Standard Error of Mean 0.76
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.071, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.4, 95% CI 2-sided [-0.17 to 2.9], Standard Error of Mean 0.76

29. Secondary Outcome: SF-36 Mental Component Summary (MCS) Score at Weeks 4, 12, 24, 36, and 52
Description: as for outcome 27
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Week 4: number analyzed (Participants) | 408 | 203 | 205 | 411
  Week 4 | 48.7 (9.73) | 46.9 (10.42) | 47.5 (10.46) | 45.5 (11.38)
  Week 12: number analyzed (Participants) | 394 | 198 | 195 | 389
  Week 12 | 49.9 (9.49) | 49.2 (9.99) | 48.8 (10.85) | 48.1 (10.26)
  Week 24: number analyzed (Participants) | 375 | 190 | 187 | 371
  Week 24 | 50.1 (9.61) | 50.1 (10.34) | 49.2 (10.11) | 49.4 (10.25)
  Week 36: number analyzed (Participants) | 348 | 178 | 179 | 327
  Week 36 | 51.1 (9.38) | 50.6 (10.26) | 49.1 (9.61) | 49.9 (10.20)
  Week 52: number analyzed (Participants) | 333 | 169 | 172 | 307
  Week 52 | 50.9 (9.32) | 50.0 (10.08) | 49.7 (10.00) | 50.2 (9.64)

30. Secondary Outcome: Change From Baseline in SF-36 MCS Score at Weeks 4, 12, 24, 36, and 52
Description: as for outcome 5
Time Frame: Baseline; Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 414 | 207 | 208 | 416
  Baseline | 44.6 (10.60) | 43.2 (11.47) | 43.1 (11.27) | 43.5 (11.50)
  Change at Week 4: number analyzed (Participants) | 406 | 203 | 203 | 411
  Change at Week 4 | 4.1 (9.32) | 3.6 (8.93) | 4.5 (9.59) | 1.9 (9.22)
  Change at Week 12: number analyzed (Participants) | 392 | 198 | 193 | 389
  Change at Week 12 | 5.3 (10.00) | 5.7 (10.04) | 5.5 (10.87) | 4.5 (10.26)
  Change at Week 24: number analyzed (Participants) | 373 | 190 | 185 | 371
  Change at Week 24 | 5.4 (10.45) | 6.6 (10.89) | 5.8 (11.26) | 6.0 (10.95)
  Change at Week 36: number analyzed (Participants) | 346 | 178 | 177 | 327
  Change at Week 36 | 6.5 (10.68) | 7.3 (11.17) | 5.4 (11.66) | 6.2 (10.96)
  Change at Week 52: number analyzed (Participants) | 331 | 169 | 170 | 307
  Change at Week 52 | 6.2 (10.74) | 6.8 (11.47) | 6.1 (11.26) | 6.5 (11.11)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.7, 95% CI 2-sided [1.6 to 3.8], Standard Error of Mean 0.57
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.032, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.5, 95% CI 2-sided [0.1 to 2.9], Standard Error of Mean 0.70
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.4, 95% CI 2-sided [1.0 to 3.8], Standard Error of Mean 0.70
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p = 0.023, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.4, 95% CI 2-sided [0.2 to 2.6], Standard Error of Mean 0.60
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p = 0.065, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.4, 95% CI 2-sided [-0.1 to 2.8], Standard Error of Mean 0.74
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.15, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.1, 95% CI 2-sided [-0.4 to 2.5], Standard Error of Mean 0.74
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.73, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.2, 95% CI 2-sided [-1.0 to 1.5], Standard Error of Mean 0.64
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.37, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.7, 95% CI 2-sided [-0.8 to 2.2], Standard Error of Mean 0.78
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.83, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-1.7 to 1.4], Standard Error of Mean 0.78
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p = 0.073, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.2, 95% CI 2-sided [-0.1 to 2.5], Standard Error of Mean 0.66
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.090, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.4, 95% CI 2-sided [-0.2 to 2.9], Standard Error of Mean 0.80
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.68, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-1.9 to 1.2], Standard Error of Mean 0.81
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.30, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.7, 95% CI 2-sided [-0.6 to 2.0], Standard Error of Mean 0.67
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.69, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.3, 95% CI 2-sided [-1.3 to 1.9], Standard Error of Mean 0.82
Statistical Analysis 15: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.95, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-1.7 to 1.5], Standard Error of Mean 0.82

31. Secondary Outcome: FACIT-Fatigue Score at Weeks 4, 12, 24, 36, and 52
Description: FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scale for a total possible score of 52.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Week 4: number analyzed (Participants) | 404 | 201 | 200 | 408
  Week 4 | 35.2 (9.82) | 34.1 (10.75) | 34.2 (10.52) | 31.4 (10.87)
  Week 12: number analyzed (Participants) | 386 | 195 | 190 | 386
  Week 12 | 38.1 (10.21) | 36.6 (11.26) | 36.9 (11.16) | 35.3 (10.23)
  Week 24: number analyzed (Participants) | 368 | 189 | 183 | 366
  Week 24 | 39.1 (10.13) | 38.7 (10.11) | 37.9 (10.76) | 37.3 (10.62)
  Week 36: number analyzed (Participants) | 345 | 177 | 177 | 324
  Week 36 | 39.8 (9.58) | 38.9 (10.19) | 38.8 (10.17) | 38.1 (9.86)
  Week 52: number analyzed (Participants) | 322 | 166 | 168 | 300
  Week 52 | 40.2 (9.36) | 38.7 (9.88) | 39.7 (10.96) | 38.4 (9.91)

32. Secondary Outcome: Change From Baseline in FACIT-Fatigue Score at Weeks 4, 12, 36, and 52
Description: as for outcome 6
Time Frame: Baseline; Weeks 4, 12, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 411 | 207 | 206 | 415
  Baseline | 28.3 (10.93) | 27.3 (11.92) | 27.3 (10.90) | 27.1 (10.72)
  Change at Week 4: number analyzed (Participants) | 403 | 201 | 198 | 408
  Change at Week 4 | 7.0 (9.46) | 6.7 (9.64) | 6.8 (9.94) | 4.3 (9.24)
  Change at Week 12: number analyzed (Participants) | 383 | 195 | 188 | 385
  Change at Week 12 | 9.8 (11.20) | 9.2 (11.21) | 9.4 (10.57) | 8.1 (10.09)
  Change at Week 36: number analyzed (Participants) | 343 | 177 | 174 | 323
  Change at Week 36 | 11.3 (11.21) | 11.9 (11.53) | 10.9 (10.81) | 11.1 (10.91)
  Change at Week 52: number analyzed (Participants) | 320 | 166 | 166 | 300
  Change at Week 52 | 11.7 (11.52) | 11.9 (12.29) | 11.5 (11.17) | 11.3 (11.49)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.2, 95% CI 2-sided [2.1 to 4.4], Standard Error of Mean 0.58
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.5, 95% CI 2-sided [1.1 to 3.9], Standard Error of Mean 0.70
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.7, 95% CI 2-sided [1.3 to 4.1], Standard Error of Mean 0.71
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.2, 95% CI 2-sided [1.0 to 3.5], Standard Error of Mean 0.64
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p = 0.13, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.2, 95% CI 2-sided [-0.4 to 2.7], Standard Error of Mean 0.78
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.032, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.7, 95% CI 2-sided [0.1 to 3.2], Standard Error of Mean 0.79
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p = 0.028, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.5, 95% CI 2-sided [0.2 to 2.8], Standard Error of Mean 0.67
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.15, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.2, 95% CI 2-sided [-0.4 to 2.7], Standard Error of Mean 0.81
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.41, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.7, 95% CI 2-sided [-0.9 to 2.3], Standard Error of Mean 0.81
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.017, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.7, 95% CI 2-sided [0.3 to 3.1], Standard Error of Mean 0.71
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.27, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.0, 95% CI 2-sided [-0.7 to 2.6], Standard Error of Mean 0.86
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.15, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.2, 95% CI 2-sided [-0.5 to 2.9], Standard Error of Mean 0.87

33. Secondary Outcome: Number of Participants by European Quality of Life 5 Dimensions (EQ-5D) Health Profile Categories at Weeks 4, 12, 24, 36, and 52
Description: The EQ-5D-5 levels (EQ-5D-5L) is a standardized measure of health status of the participant at the visit (same day) that provides a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L consists of 2 components: a descriptive system of the participant's health and a rating of his or her current health state on a 0-100 VAS. The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Rating gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
Participants
  Mobility: Week 4: number analyzed (Participants) | 406 | 202 | 201 | 410
  Mobility: Week 4: No Problems | 161 | 66 | 81 | 104
  Mobility: Week 4: Slight Problems | 149 | 68 | 56 | 135
  Mobility: Week 4: Moderate Problems | 82 | 50 | 38 | 116
  Mobility: Week 4: Severe Problems | 13 | 17 | 20 | 54
  Mobility: Week 4: Extreme Problems | 1 | 1 | 6 | 1
  Mobility: Week 12: number analyzed (Participants) | 390 | 196 | 192 | 388
  Mobility: Week 12: No Problems | 198 | 87 | 86 | 138
  Mobility: Week 12: Slight Problems | 135 | 56 | 60 | 135
  Mobility: Week 12: Moderate Problems | 41 | 36 | 27 | 91
  Mobility: Week 12: Severe Problems | 12 | 17 | 14 | 20
  Mobility: Week 12: Extreme Problems | 4 | 0 | 5 | 4
  Mobility: Week 24: number analyzed (Participants) | 377 | 192 | 184 | 370
  Mobility: Week 24: No Problems | 208 | 92 | 95 | 152
  Mobility: Week 24: Slight Problems | 116 | 55 | 50 | 135
  Mobility: Week 24: Moderate Problems | 46 | 36 | 24 | 63
  Mobility: Week 24: Severe Problems | 5 | 9 | 13 | 16
  Mobility: Week 24: Extreme Problems | 2 | 0 | 2 | 4
  Mobility: Week 36: number analyzed (Participants) | 365 | 188 | 180 | 356
  Mobility: Week 36: No Problems | 216 | 93 | 98 | 152
  Mobility: Week 36: Slight Problems | 96 | 60 | 46 | 135
  Mobility: Week 36: Moderate Problems | 48 | 30 | 27 | 51
  Mobility: Week 36: Severe Problems | 5 | 5 | 8 | 16
  Mobility: Week 36: Extreme Problems | 0 | 0 | 1 | 2
  Mobility: Week 52: number analyzed (Participants) | 347 | 176 | 174 | 334
  Mobility: Week 52: No Problems | 217 | 91 | 93 | 156
  Mobility: Week 52: Slight Problems | 92 | 50 | 47 | 108
  Mobility: Week 52: Moderate Problems | 28 | 29 | 21 | 54
  Mobility: Week 52: Severe Problems | 9 | 6 | 10 | 15
  Mobility: Week 52: Extreme Problems | 1 | 0 | 3 | 1
  Self-Care: Week 4: number analyzed (Participants) | 406 | 202 | 201 | 410
  Self-Care: Week 4: No Problems | 214 | 99 | 102 | 143
  Self-Care: Week 4: Slight Problems | 142 | 63 | 50 | 141
  Self-Care: Week 4: Moderate Problems | 42 | 28 | 38 | 96
  Self-Care: Week 4: Severe Problems | 7 | 9 | 10 | 29
  Self-Care: Week 4: Extreme Problems | 1 | 3 | 1 | 1
  Self-Care: Week 12: number analyzed (Participants) | 390 | 196 | 192 | 388
  Self-Care: Week 12: No Problems | 277 | 113 | 111 | 190
  Self-Care: Week 12: Slight Problems | 85 | 55 | 55 | 129
  Self-Care: Week 12: Moderate Problems | 19 | 22 | 21 | 54
  Self-Care: Week 12: Severe Problems | 6 | 5 | 4 | 13
  Self-Care: Week 12: Extreme Problems | 3 | 1 | 1 | 2
  Self-Care: Week 24: number analyzed (Participants) | 377 | 192 | 184 | 370
  Self-Care: Week 24: No Problems | 283 | 128 | 112 | 222
  Self-Care: Week 24: Slight Problems | 73 | 42 | 52 | 95
  Self-Care: Week 24: Moderate Problems | 16 | 20 | 17 | 46
  Self-Care: Week 24: Severe Problems | 1 | 2 | 3 | 5
  Self-Care: Week 24: Extreme Problems | 4 | 0 | 0 | 2
  Self-Care: Week 36: number analyzed (Participants) | 365 | 188 | 180 | 356
  Self-Care: Week 36: No Problems | 271 | 122 | 121 | 224
  Self-Care: Week 36: Slight Problems | 70 | 44 | 41 | 93
  Self-Care: Week 36: Moderate Problems | 20 | 21 | 16 | 31
  Self-Care: Week 36: Severe Problems | 3 | 1 | 1 | 5
  Self-Care: Week 36: Extreme Problems | 1 | 0 | 1 | 3
  Self-Care: Week 52: number analyzed (Participants) | 347 | 176 | 174 | 334
  Self-Care: Week 52: No Problems | 268 | 117 | 117 | 208
  Self-Care: Week 52: Slight Problems | 60 | 36 | 36 | 84
  Self-Care: Week 52: Moderate Problems | 13 | 21 | 16 | 35
  Self-Care: Week 52: Severe Problems | 5 | 2 | 4 | 6
  Self-Care: Week 52: Extreme Problems | 1 | 0 | 1 | 1
  Usual Activities: Week 4: number analyzed (Participants) | 406 | 202 | 201 | 410
  Usual Activities: Week 4: No Problems | 118 | 50 | 54 | 80
  Usual Activities: Week 4: Slight Problems | 180 | 86 | 81 | 153
  Usual Activities: Week 4: Moderate Problems | 90 | 47 | 49 | 122
  Usual Activities: Week 4: Severe Problems | 16 | 19 | 14 | 49
  Usual Activities: Week 4: Extreme Problems | 2 | 0 | 3 | 6
  Usual Activities: Week 12: number analyzed (Participants) | 390 | 196 | 192 | 388
  Usual Activities: Week 12: No Problems | 185 | 78 | 83 | 101
  Usual Activities: Week 12: Slight Problems | 148 | 65 | 61 | 179
  Usual Activities: Week 12: Moderate Problems | 44 | 42 | 35 | 85
  Usual Activities: Week 12: Severe Problems | 11 | 9 | 11 | 19
  Usual Activities: Week 12: Extreme Problems | 2 | 2 | 2 | 4
  Usual Activities: Week 24: number analyzed (Participants) | 377 | 192 | 184 | 370
  Usual Activities: Week 24: No Problems | 188 | 92 | 83 | 142
  Usual Activities: Week 24: Slight Problems | 135 | 60 | 63 | 147
  Usual Activities: Week 24: Moderate Problems | 43 | 31 | 30 | 64
  Usual Activities: Week 24: Severe Problems | 8 | 9 | 8 | 13
  Usual Activities: Week 24: Extreme Problems | 3 | 0 | 0 | 4
  Usual Activities: Week 36: number analyzed (Participants) | 365 | 188 | 180 | 356
  Usual Activities: Week 36: No Problems | 199 | 86 | 92 | 158
  Usual Activities: Week 36: Slight Problems | 119 | 61 | 51 | 134
  Usual Activities: Week 36: Moderate Problems | 42 | 37 | 31 | 50
  Usual Activities: Week 36: Severe Problems | 5 | 4 | 3 | 12
  Usual Activities: Week 36: Extreme Problems | 0 | 0 | 3 | 2
  Usual Activities: Week 52: number analyzed (Participants) | 347 | 176 | 174 | 334
  Usual Activities: Week 52: No Problems | 203 | 84 | 92 | 147
  Usual Activities: Week 52: Slight Problems | 106 | 62 | 48 | 125
  Usual Activities: Week 52: Moderate Problems | 31 | 22 | 27 | 50
  Usual Activities: Week 52: Severe Problems | 7 | 7 | 5 | 10
  Usual Activities: Week 52: Extreme Problems | 0 | 1 | 2 | 2
  Pain/Discomfort: Week 4: number analyzed (Participants) | 406 | 202 | 201 | 410
  Pain/Discomfort: Week 4: No Problems | 45 | 23 | 21 | 18
  Pain/Discomfort: Week 4: Slight Problems | 208 | 85 | 91 | 131
  Pain/Discomfort: Week 4: Moderate Problems | 132 | 73 | 60 | 173
  Pain/Discomfort: Week 4: Severe Problems | 21 | 19 | 26 | 78
  Pain/Discomfort: Week 4: Extreme Problems | 0 | 2 | 3 | 10
  Pain/Discomfort: Week 12: number analyzed (Participants) | 390 | 196 | 192 | 388
  Pain/Discomfort: Week 12: No Problems | 93 | 35 | 38 | 41
  Pain/Discomfort: Week 12: Slight Problems | 202 | 96 | 81 | 167
  Pain/Discomfort: Week 12: Moderate Problems | 83 | 47 | 53 | 143
  Pain/Discomfort: Week 12: Severe Problems | 12 | 15 | 16 | 35
  Pain/Discomfort: Week 12: Extreme Problems | 0 | 3 | 4 | 2
  Pain/Discomfort: Week 24: number analyzed (Participants) | 377 | 192 | 184 | 370
  Pain/Discomfort: Week 24: No Problems | 110 | 46 | 40 | 44
  Pain/Discomfort: Week 24: Slight Problems | 182 | 91 | 93 | 206
  Pain/Discomfort: Week 24: Moderate Problems | 75 | 46 | 42 | 98
  Pain/Discomfort: Week 24: Severe Problems | 9 | 9 | 7 | 22
  Pain/Discomfort: Week 24: Extreme Problems | 1 | 0 | 2 | 0
  Pain/Discomfort: Week 36: number analyzed (Participants) | 365 | 188 | 180 | 356
  Pain/Discomfort: Week 36: No Problems | 102 | 43 | 39 | 57
  Pain/Discomfort: Week 36: Slight Problems | 188 | 90 | 87 | 195
  Pain/Discomfort: Week 36: Moderate Problems | 68 | 41 | 44 | 85
  Pain/Discomfort: Week 36: Severe Problems | 6 | 14 | 7 | 18
  Pain/Discomfort: Week 36: Extreme Problems | 1 | 0 | 3 | 1
  Pain/Discomfort: Week 52: number analyzed (Participants) | 347 | 176 | 174 | 334
  Pain/Discomfort: Week 52: No Problems | 108 | 46 | 49 | 63
  Pain/Discomfort: Week 52: Slight Problems | 169 | 82 | 88 | 168
  Pain/Discomfort: Week 52: Moderate Problems | 59 | 40 | 25 | 80
  Pain/Discomfort: Week 52: Severe Problems | 11 | 8 | 9 | 22
  Pain/Discomfort: Week 52: Extreme Problems | 0 | 0 | 3 | 1
  Anxiety/Depression: Week 4: number analyzed (Participants) | 406 | 202 | 201 | 410
  Anxiety/Depression: Week 4: No Problems | 221 | 101 | 94 | 159
  Anxiety/Depression: Week 4: Slight Problems | 126 | 58 | 64 | 148
  Anxiety/Depression: Week 4: Moderate Problems | 53 | 33 | 35 | 73
  Anxiety/Depression: Week 4: Severe Problems | 6 | 10 | 6 | 25
  Anxiety/Depression: Week 4: Extreme Problems | 0 | 0 | 2 | 5
  Anxiety/Depression: Week 12: number analyzed (Participants) | 390 | 196 | 192 | 388
  Anxiety/Depression: Week 12: No Problems | 233 | 104 | 106 | 198
  Anxiety/Depression: Week 12: Slight Problems | 114 | 62 | 58 | 125
  Anxiety/Depression: Week 12: Moderate Problems | 28 | 19 | 17 | 49
  Anxiety/Depression: Week 12: Severe Problems | 14 | 9 | 10 | 15
  Anxiety/Depression: Week 12: Extreme Problems | 1 | 2 | 1 | 1
  Anxiety/Depression: Week 24: number analyzed (Participants) | 377 | 192 | 184 | 370
  Anxiety/Depression: Week 24: No Problems | 236 | 117 | 103 | 219
  Anxiety/Depression: Week 24: Slight Problems | 97 | 47 | 64 | 93
  Anxiety/Depression: Week 24: Moderate Problems | 32 | 25 | 11 | 42
  Anxiety/Depression: Week 24: Severe Problems | 9 | 3 | 6 | 14
  Anxiety/Depression: Week 24: Extreme Problems | 3 | 0 | 0 | 2
  Anxiety/Depression: Week 36: number analyzed (Participants) | 365 | 188 | 180 | 356
  Anxiety/Depression: Week 36: No Problems | 233 | 119 | 103 | 194
  Anxiety/Depression: Week 36: Slight Problems | 99 | 50 | 56 | 116
  Anxiety/Depression: Week 36: Moderate Problems | 31 | 13 | 17 | 32
  Anxiety/Depression: Week 36: Severe Problems | 2 | 5 | 3 | 12
  Anxiety/Depression: Week 36: Extreme Problems | 0 | 1 | 1 | 2
  Anxiety/Depression: Week 52: number analyzed (Participants) | 347 | 176 | 174 | 334
  Anxiety/Depression: Week 52: No Problems | 222 | 113 | 106 | 182
  Anxiety/Depression: Week 52: Slight Problems | 94 | 40 | 43 | 100
  Anxiety/Depression: Week 52: Moderate Problems | 26 | 18 | 20 | 45
  Anxiety/Depression: Week 52: Severe Problems | 5 | 5 | 3 | 5
  Anxiety/Depression: Week 52: Extreme Problems | 0 | 0 | 2 | 2

34. Secondary Outcome: EQ-5D Current Health VAS at Weeks 4, 12, 24, 36, and 52
Description: EQ-5D-5L is a standardized measure of health status of the participant at the visit (same day) that provides a simple, generic measure of health for clinical and economic appraisal. Participant rates their current health state on a 0-100 VAS. It gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Week 4: number analyzed (Participants) | 404 | 201 | 200 | 408
  Week 4 | 65 (18.7) | 61 (21.6) | 62 (20.0) | 56 (21.2)
  Week 12: number analyzed (Participants) | 386 | 195 | 190 | 386
  Week 12 | 69 (21.3) | 67 (22.9) | 66 (22.7) | 64 (20.7)
  Week 24: number analyzed (Participants) | 368 | 189 | 183 | 366
  Week 24 | 73 (21.0) | 72 (19.6) | 68 (22.4) | 69 (21.3)
  Week 36: number analyzed (Participants) | 344 | 177 | 177 | 324
  Week 36 | 73 (22.1) | 71 (21.8) | 69 (21.1) | 68 (22.8)
  Week 52: number analyzed (Participants) | 322 | 166 | 168 | 300
  Week 52 | 75 (21.7) | 72 (22.1) | 71 (23.7) | 71 (21.2)

35. Secondary Outcome: Change From Baseline in EQ-5D Current Health VAS at Weeks 4, 12, 24, 36, and 52
Description: The EQ-5D-5L is a standardized measure of health status of the participant at the visit (same day) that provides a simple, generic measure of health for clinical and economic appraisal. Participant rates their current health state on a 0-100 VAS. It gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health. Positive change indicates improvement (better health).
Time Frame: Baseline; Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
score on a scale
  Baseline: number analyzed (Participants) | 411 | 207 | 206 | 415
  Baseline | 50 (22.0) | 50 (24.6) | 51 (22.5) | 50 (22.1)
  Change at Week 4: number analyzed (Participants) | 403 | 201 | 198 | 408
  Change at Week 4 | 16 (25.0) | 10 (24.6) | 11 (22.4) | 7 (25.0)
  Change at Week 12: number analyzed (Participants) | 383 | 195 | 188 | 385
  Change at Week 12 | 19 (29.8) | 17 (28.0) | 15 (26.1) | 14 (27.7)
  Change at Week 24: number analyzed (Participants) | 365 | 189 | 181 | 365
  Change at Week 24 | 24 (28.1) | 21 (27.7) | 17 (29.0) | 19 (28.8)
  Change at Week 36: number analyzed (Participants) | 342 | 177 | 174 | 323
  Change at Week 36 | 23 (29.7) | 21 (28.6) | 18 (28.8) | 19 (29.8)
  Change at Week 52: number analyzed (Participants) | 320 | 166 | 166 | 300
  Change at Week 52 | 26 (31.1) | 22 (31.5) | 20 (30.1) | 22 (30.6)
Statistical Analysis 1: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 4]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 9.0, 95% CI 2-sided [6.0 to 12.0], Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 4.0, 95% CI 2-sided [1.0 to 8.0], Standard Error of Mean 1.6
Statistical Analysis 3: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 6.0, 95% CI 2-sided [3.0 to 9.0], Standard Error of Mean 1.6
Statistical Analysis 4: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 7]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 5.0, 95% CI 2-sided [2.0 to 8.0], Standard Error of Mean 1.5
Statistical Analysis 5: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 8]; Test type: Superiority; p = 0.089, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.0, 95% CI 2-sided [-0.0 to 7.0], Standard Error of Mean 1.8
Statistical Analysis 6: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 9]; Test type: Superiority; p = 0.18, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.0, 95% CI 2-sided [-1.0 to 6.0], Standard Error of Mean 1.9
Statistical Analysis 7: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 4.0, 95% CI 2-sided [1.0 to 7.0], Standard Error of Mean 1.5
Statistical Analysis 8: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.049, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 4.0, 95% CI 2-sided [0.0 to 7.0], Standard Error of Mean 1.8
Statistical Analysis 9: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.84, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.0, 95% CI 2-sided [-4.0 to 3.0], Standard Error of Mean 1.8
Statistical Analysis 10: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 6.0, 95% CI 2-sided [2.0 to 9.0], Standard Error of Mean 1.6
Statistical Analysis 11: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 11, analysis 11]; Test type: Superiority; p = 0.078, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.0, 95% CI 2-sided [-0.0 to 7.0], Standard Error of Mean 2.0
Statistical Analysis 12: Comparison: Filgotinib 200 mg Monotherapy vs MTX Monotherapy; [analysis description as in outcome 11, analysis 12]; Test type: Superiority; p = 0.39, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.0, 95% CI 2-sided [-2.0 to 6.0], Standard Error of Mean 2.0
Statistical Analysis 13: Comparison: Filgotinib 200 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.004, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 5.0, 95% CI 2-sided [2.0 to 8.0], Standard Error of Mean 1.7
Statistical Analysis 14: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 2]; Test type: Superiority; p = 0.45, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.0, 95% CI 2-sided [-3.0 to 6.0], Standard Error of Mean 2.1
Statistical Analysis 15: Comparison: Filgotinib 100 mg + MTX vs MTX Monotherapy; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.85, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.0, 95% CI 2-sided [-4.0 to 5.0], Standard Error of Mean 2.1

36. Secondary Outcome: Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA): Mean Percentage of Work Time Missed (Absenteeism) at Weeks 4, 12, 24, 36, and 52
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: currently employed; work time missed due to RA; work time missed due to other reasons; hours actually worked; degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages. Higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of work time missed
  Week 4: number analyzed (Participants) | 167 | 77 | 87 | 150
  Week 4 | 10.1 (23.95) | 15.4 (30.46) | 9.2 (21.88) | 16.0 (30.49)
  Week 12: number analyzed (Participants) | 163 | 72 | 84 | 161
  Week 12 | 6.7 (19.11) | 7.3 (18.29) | 12.6 (24.42) | 11.3 (25.59)
  Week 24: number analyzed (Participants) | 164 | 72 | 86 | 145
  Week 24 | 6.4 (19.93) | 5.7 (13.96) | 12.4 (23.14) | 5.1 (14.21)
  Week 36: number analyzed (Participants) | 156 | 73 | 85 | 131
  Week 36 | 5.5 (15.78) | 7.0 (17.90) | 11.5 (25.28) | 5.6 (16.90)
  Week 52: number analyzed (Participants) | 149 | 69 | 76 | 120
  Week 52 | 4.6 (14.62) | 8.5 (20.70) | 9.8 (22.21) | 6.4 (19.84)

37. Secondary Outcome: WPAI-RA: Mean Percentage of Impairment While Working Due to RA (Presenteeism) at Weeks 4, 12, 24, 36, and 52
Description: as for outcome 36
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of impairment while working
  Week 4: number analyzed (Participants) | 160 | 70 | 84 | 137
  Week 4 | 29.6 (24.21) | 29.4 (27.76) | 33.9 (24.10) | 45.3 (26.04)
  Week 12: number analyzed (Participants) | 160 | 72 | 81 | 152
  Week 12 | 22.6 (23.43) | 23.6 (24.85) | 26.0 (24.78) | 32.5 (24.31)
  Week 24: number analyzed (Participants) | 160 | 72 | 84 | 144
  Week 24 | 17.9 (18.95) | 18.1 (19.40) | 23.2 (24.70) | 23.3 (21.18)
  Week 36: number analyzed (Participants) | 155 | 72 | 81 | 129
  Week 36 | 15.5 (18.38) | 16.3 (20.31) | 20.9 (24.04) | 22.7 (24.10)
  Week 52: number analyzed (Participants) | 148 | 67 | 74 | 116
  Week 52 | 14.5 (18.08) | 19.6 (22.32) | 16.5 (23.08) | 18.3 (16.95)

38. Secondary Outcome: WPAI-RA: Mean Percentage of Overall Work Productivity Impairment Due to RA at Weeks 4, 12, 24, 36, and 52
Description: as for outcome 36
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of overall work productivity
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of overall work productivity
  Week 4: number analyzed (Participants) | 160 | 70 | 84 | 137
  Week 4 | 32.8 (25.79) | 32.3 (29.18) | 37.0 (25.87) | 48.6 (27.40)
  Week 12: number analyzed (Participants) | 160 | 72 | 81 | 152
  Week 12 | 25.1 (26.42) | 26.7 (28.11) | 31.4 (28.43) | 35.5 (26.13)
  Week 24: number analyzed (Participants) | 160 | 72 | 84 | 144
  Week 24 | 20.2 (22.36) | 22.4 (22.92) | 29.3 (28.98) | 26.2 (23.45)
  Week 36: number analyzed (Participants) | 155 | 72 | 81 | 129
  Week 36 | 18.8 (22.09) | 20.9 (23.34) | 24.5 (28.11) | 25.0 (25.89)
  Week 52: number analyzed (Participants) | 148 | 67 | 74 | 116
  Week 52 | 17.2 (21.61) | 22.9 (25.21) | 21.2 (27.26) | 20.7 (18.67)

39. Secondary Outcome: WPAI-RA: Mean Percentage of Activity Impairment Due to RA at Weeks 4, 12, 24, 36, and 52
Description: as for outcome 36
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of activity impairment
  Week 4: number analyzed (Participants) | 404 | 201 | 200 | 408
  Week 4 | 40.4 (25.52) | 46.8 (27.82) | 45.4 (25.65) | 51.6 (24.73)
  Week 12: number analyzed (Participants) | 386 | 195 | 190 | 386
  Week 12 | 30.6 (25.53) | 36.1 (26.77) | 34.7 (27.29) | 41.1 (24.75)
  Week 24: number analyzed (Participants) | 368 | 189 | 183 | 366
  Week 24 | 26.5 (23.32) | 29.5 (26.02) | 32.3 (26.92) | 32.1 (24.44)
  Week 36: number analyzed (Participants) | 344 | 177 | 177 | 324
  Week 36 | 23.5 (22.54) | 29.7 (27.03) | 29.0 (26.08) | 31.8 (25.55)
  Week 52: number analyzed (Participants) | 322 | 166 | 168 | 300
  Week 52 | 22.5 (22.80) | 28.2 (26.54) | 25.6 (25.19) | 28.8 (23.81)

40. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Work Time Missed (Absenteeism) at Weeks 4, 12, 24, 36, and 52
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: currently employed; work time missed due to RA; work time missed due to other reasons; hours actually worked; degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages, higher numbers indicate greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of work time missed
  Baseline: number analyzed (Participants) | 171 | 78 | 88 | 167
  Baseline | 12.8 (24.29) | 20.1 (32.36) | 13.5 (26.35) | 15.6 (28.79)
  Change at Week 4: number analyzed (Participants) | 155 | 70 | 82 | 138
  Change at Week 4 | -1.5 (25.68) | -3.3 (24.44) | -4.0 (21.08) | -1.3 (23.73)
  Change at Week 12: number analyzed (Participants) | 142 | 67 | 75 | 141
  Change at Week 12 | -4.9 (25.11) | -11.0 (32.65) | -2.3 (23.52) | -5.2 (29.01)
  Change at Week 24: number analyzed (Participants) | 141 | 63 | 77 | 122
  Change at Week 24 | -4.8 (28.91) | -15.5 (34.51) | -3.1 (28.77) | -10.6 (29.08)
  Change at Week 36: number analyzed (Participants) | 130 | 62 | 69 | 107
  Change at Week 36 | -6.7 (28.20) | -16.4 (35.63) | -4.1 (26.83) | -7.9 (29.99)
  Change at Week 52: number analyzed (Participants) | 124 | 59 | 65 | 97
  Change at Week 52 | -4.8 (23.27) | -15.7 (32.72) | -2.8 (29.12) | -6.7 (31.63)

41. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Impairment While Working Due to RA (Presenteeism) at Weeks 4, 12, 24, 36, and 52
Description: as for outcome 40
Time Frame: Baseline; Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of impairment while working
  Baseline: number analyzed (Participants) | 163 | 70 | 82 | 154
  Baseline | 47.3 (26.32) | 49.0 (28.45) | 52.1 (25.81) | 53.6 (27.12)
  Change at Week 4: number analyzed (Participants) | 144 | 62 | 77 | 125
  Change at Week 4 | -17.8 (25.34) | -19.8 (27.49) | -18.3 (28.58) | -7.4 (20.55)
  Change at Week 12: number analyzed (Participants) | 135 | 61 | 70 | 126
  Change at Week 12 | -25.6 (27.09) | -28.4 (29.39) | -26.0 (24.70) | -20.7 (27.83)
  Change at Week 24: number analyzed (Participants) | 132 | 56 | 72 | 113
  Change at Week 24 | -27.1 (26.77) | -32.9 (28.20) | -27.9 (27.06) | -28.3 (29.06)
  Change at Week 36: number analyzed (Participants) | 123 | 55 | 64 | 99
  Change at Week 36 | -29.1 (24.99) | -33.8 (27.99) | -30.3 (29.38) | -28.8 (31.92)
  Change at Week 52: number analyzed (Participants) | 120 | 51 | 61 | 89
  Change at Week 52 | -32.3 (26.81) | -32.7 (31.75) | -33.3 (29.25) | -31.5 (28.23)

42. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Overall Work Productivity Impairment Due to RA at Weeks 4, 12, 24, 36, and 52
Description: as for outcome 40
Time Frame: Baseline; Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of overall work productivity
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of overall work productivity
  Baseline: number analyzed (Participants) | 163 | 70 | 82 | 154
  Baseline | 50.8 (27.28) | 51.6 (30.10) | 54.4 (25.60) | 56.1 (28.00)
  Change at Week 4: number analyzed (Participants) | 144 | 62 | 77 | 125
  Change at Week 4 | -17.6 (26.21) | -19.0 (29.43) | -17.6 (28.69) | -6.4 (22.27)
  Change at Week 12: number analyzed (Participants) | 135 | 61 | 70 | 126
  Change at Week 12 | -26.3 (28.85) | -27.5 (30.53) | -23.5 (26.01) | -20.1 (28.63)
  Change at Week 24: number analyzed (Participants) | 132 | 56 | 72 | 113
  Change at Week 24 | -28.5 (27.71) | -31.3 (30.04) | -24.7 (29.61) | -27.9 (29.31)
  Change at Week 36: number analyzed (Participants) | 123 | 55 | 64 | 99
  Change at Week 36 | -29.3 (26.76) | -33.1 (31.56) | -29.1 (31.79) | -29.2 (32.72)
  Change at Week 52: number analyzed (Participants) | 120 | 51 | 61 | 89
  Change at Week 52 | -33.0 (28.74) | -33.5 (32.34) | -30.6 (31.24) | -30.8 (28.76)

43. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Activity Impairment Due to RA at Weeks 4, 12, 24, 36, and 52
Description: as for outcome 40
Time Frame: Baseline; Weeks 4, 12, 24, 36, and 52
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
Number analyzed (Participants) | 416 | 207 | 210 | 416
percentage of activity impairment
  Baseline: number analyzed (Participants) | 411 | 207 | 206 | 415
  Baseline | 60.2 (23.36) | 62.8 (23.10) | 63.3 (24.37) | 64.0 (22.59)
  Change at Week 4: number analyzed (Participants) | 403 | 201 | 198 | 408
  Change at Week 4 | -19.9 (24.07) | -15.8 (23.90) | -17.8 (27.11) | -12.4 (23.80)
  Change at Week 12: number analyzed (Participants) | 383 | 195 | 188 | 385
  Change at Week 12 | -29.4 (27.15) | -26.4 (26.19) | -28.7 (27.80) | -22.7 (25.32)
  Change at Week 24: number analyzed (Participants) | 365 | 189 | 181 | 365
  Change at Week 24 | -33.1 (26.84) | -33.2 (26.97) | -31.2 (28.01) | -31.5 (27.80)
  Change at Week 36: number analyzed (Participants) | 342 | 177 | 174 | 323
  Change at Week 36 | -35.6 (26.52) | -33.8 (26.48) | -34.1 (28.26) | -32.1 (28.47)
  Change at Week 52: number analyzed (Participants) | 320 | 166 | 166 | 300
  Change at Week 52 | -36.7 (27.11) | -35.4 (28.32) | -36.7 (28.37) | -34.2 (28.83)

ADVERSE EVENTS:
Time Frame: First dose date up to last dose date (Maximum: 56 weeks) plus 30 days
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Filgotinib 200 mg + MTX: Participants were administered filgotinib 200 mg orally, once daily + placebo to match (PTM) filgotinib 100 mg orally, once daily + methotrexate (MTX) up to 20 mg orally, once weekly for up to 54 weeks.
Arm/Group | Filgotinib 200 mg + MTX | Filgotinib 100 mg + MTX | Filgotinib 200 mg Monotherapy | MTX Monotherapy
All-Cause Mortality (participants affected / at risk) | 3/416 | 1/207 | 0/210 | 0/416
Serious Adverse Events (participants affected / at risk) | 26/416 | 13/207 | 17/210 | 28/416
Other Adverse Events (participants affected / at risk) | 179/416 | 88/207 | 78/210 | 164/416
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg + MTX (N=416) | Filgotinib 100 mg + MTX (N=207) | Filgotinib 200 mg Monotherapy (N=210) | MTX Monotherapy (N=416)
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Lupus myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0
Abdominal hernia infection (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia cryptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Pyonephrosis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Giant cell tumour of tendon sheath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral amyloid angiopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Vertebral artery aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Rheumatoid vasculitis (Vascular disorders) | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg + MTX (N=416) | Filgotinib 100 mg + MTX (N=207) | Filgotinib 200 mg Monotherapy (N=210) | MTX Monotherapy (N=416)
Diarrhoea (Gastrointestinal disorders) | 17 | 12 | 6 | 21
Nausea (Gastrointestinal disorders) | 51 | 35 | 15 | 50
Bronchitis (Infections and infestations) | 12 | 11 | 4 | 15
Nasopharyngitis (Infections and infestations) | 21 | 17 | 17 | 25
Upper respiratory tract infection (Infections and infestations) | 42 | 9 | 14 | 34
Urinary tract infection (Infections and infestations) | 19 | 13 | 11 | 11
Alanine aminotransferase increased (Investigations) | 23 | 6 | 3 | 11
Headache (Nervous system disorders) | 23 | 8 | 8 | 25
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 15 | 4 | 20
Hypertension (Vascular disorders) | 21 | 10 | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT02886728/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT02886728/SAP_001.pdf